CLINICAL TRIAL: NCT00474526
Title: A Phase 3, Open-Label, Randomized, Parallel-Group, Multi-Center Study to Evaluate the Safety and Immunogenicity of Novartis Meningococcal ACWY Conjugate Vaccine When Administered With Routine Infant Vaccinations to Healthy Infants
Brief Title: A Study to Evaluate Safety and Immune Response of Novartis Meningococcal ACWY Vaccine In Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V59P14
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Results first posted 2014-03-24 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-02

CONDITIONS: Meningitis, Meningococcal
Keywords: Meningococcal; meningitis; vaccine; infants; Meningococcal meningitis; Meningococcal disease
MeSH Terms: conditions — Meningitis, Meningococcal; Meningitis; Meningococcal Infections | interventions — Meningococcal Vaccines; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; PEDIARIX; Tetanus Toxoid; Hepatitis B Vaccines; Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate; Pneumococcal Vaccines; Heptavalent Pneumococcal Conjugate Vaccine; Hepatitis A Vaccines; measles, mumps, rubella, varicella vaccine; Chickenpox Vaccine; Diphtheria-Tetanus-acellular Pertussis Vaccines

ARMS (17):
- US1A (MenACWY-CRM + Infant Vaccines) (Experimental): Received vaccines:
  MenACWY: 2, 4, 6, and 12 months
  DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines: 2, 4, and 6 months
  Pneumococcal, HAV, and MMR-V: 12 months
  Interventions: Biological: Meningococcal ACWY Conjugate Vaccine; Biological: DTaP-IPV-HBV; Biological: Hib; Biological: Rotavirus; Biological: Pneumococcal 7-valent Conjugate Vaccine; Biological: HAV; Biological: MMR-V
- US1B (MenACWY-CRM + Infant Vaccines) (Experimental): Received vaccines:
  MenACWY: 2, 4, 6, and 13 months
  DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines: 2, 4, and 6 months
  Pneumococcal, HAV, and MMR-V: 12 months
  Interventions: Biological: Meningococcal ACWY Conjugate Vaccine; Biological: DTaP-IPV-HBV; Biological: Hib; Biological: Rotavirus; Biological: Pneumococcal 7-valent Conjugate Vaccine; Biological: HAV; Biological: MMR-V
- US2 (Infant Vaccines Only) (Experimental): Received vaccines:
  MenACWY: 12 and 15 months
  DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines: 2, 4, and 6 months
  Pneumococcal, HAV, and MMR-V: 12 months
  Interventions: Biological: Meningococcal ACWY Conjugate Vaccine; Biological: DTaP-IPV-HBV; Biological: Hib; Biological: Rotavirus; Biological: Pneumococcal 7-valent Conjugate Vaccine; Biological: HAV; Biological: MMR-V
- US3 (MenACWY-CRM + Infant Vaccines) (Experimental): Received vaccines:
  MenACWY: 2, 4, 6, and 12 months
  DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines: 2, 4, and 6 months
  Pneumococcal, HAV, and MMR-V: 12 months
  Interventions: Biological: Meningococcal ACWY Conjugate Vaccine; Biological: DTaP-IPV-HBV; Biological: Hib; Biological: Rotavirus; Biological: Pneumococcal 7-valent Conjugate Vaccine; Biological: HAV; Biological: MMR-V
- US4A (Infant Vaccines Only) (Experimental): Received vaccines:
  MenACWY: 12 and 15 months
  DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines: 2, 4, and 6 months
  Pneumococcal, HAV, and MMR-V: 12 months
  Interventions: Biological: Meningococcal ACWY Conjugate Vaccine; Biological: DTaP-IPV-HBV; Biological: Hib; Biological: Rotavirus; Biological: HAV; Biological: MMR-V
- US4B (Infant Vaccines Only) (Experimental): Received vaccines:
  MenACWY: 13 and 15 months DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines: 2, 4, and 6 months
  Pneumococcal, HAV, and MMR-V: 12 months
  Interventions: Biological: Meningococcal ACWY Conjugate Vaccine; Biological: DTaP-IPV-HBV; Biological: Hib; Biological: Rotavirus; Biological: Pneumococcal 7-valent Conjugate Vaccine; Biological: HAV; Biological: MMR-V
- US4C (Infant Vaccines Only) (Experimental): Received vaccines:
  MenACWY: 18 months
  DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines: 2, 4, and 6 months
  Pneumococcal, HAV, and MMR-V: 12 months
  Interventions: Biological: Meningococcal ACWY Conjugate Vaccine; Biological: DTaP-IPV-HBV; Biological: Hib; Biological: Rotavirus; Biological: Pneumococcal 7-valent Conjugate Vaccine; Biological: HAV; Biological: MMR-V
- LA1A (MenACWY-CRM + Infant Vaccines) (Experimental): Received vaccines:
  MenACWY: 2, 6, and 12 months
  DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines: 2, 4, and 6 months Pneumococcal, HAV, and MMR-V: 12 months
  Interventions: Biological: Meningococcal ACWY Conjugate Vaccine; Biological: DTaP-IPV-HBV; Biological: Hib; Biological: Rotavirus; Biological: Pneumococcal 7-valent Conjugate Vaccine; Biological: HAV; Biological: MMR-V
- LA1B (MenACWY-CRM + Infant Vaccines) (Experimental): Received vaccines:
  MenACWY: 2, 6, and 13 months
  DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines: 2, 4, and 6 months
  Pneumococcal, HAV, and MMR-V: 12 months
  Interventions: Biological: Meningococcal ACWY Conjugate Vaccine; Biological: DTaP-IPV-HBV; Biological: Hib; Biological: Rotavirus; Biological: Pneumococcal 7-valent Conjugate Vaccine; Biological: HAV; Biological: MMR-V
- LA2 (Infant Vaccines Only) (Experimental): Received vaccines:
  MenACWY: 12 and 15 months
  DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines: 2, 4, and 6 months
  Pneumococcal, HAV, and MMR-V: 12 months
  Interventions: Biological: Meningococcal ACWY Conjugate Vaccine; Biological: DTaP-IPV-HBV; Biological: Hib; Biological: Rotavirus; Biological: Pneumococcal 7-valent Conjugate Vaccine; Biological: HAV; Biological: MMR-V
- LA3A (MenACWY-CRM + Infant Vaccines) (Experimental): Received vaccines:
  MenACWY: 2, 4, 6, and 16 months
  DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines: 2, 4, and 6 months
  DTaP, Hib: 16 months
  Pneumococcal, HAV, and MMR-V: 12 months
  Interventions: Biological: Meningococcal ACWY Conjugate Vaccine; Biological: DTaP-IPV-HBV; Biological: Hib; Biological: Rotavirus; Biological: Pneumococcal 7-valent Conjugate Vaccine; Biological: HAV; Biological: MMR-V; Biological: DTaP
- LA3B (MenACWY-CRM + Infant Vaccines) (Experimental): Received vaccines:
  MenACWY: 2, 4, 6, and 17 months
  DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines: 2, 4, and 6 months
  DTaP, Hib: 16 months
  Pneumococcal, HAV, and MMR-V: 12 months
  Interventions: Biological: Meningococcal ACWY Conjugate Vaccine; Biological: DTaP-IPV-HBV; Biological: Hib; Biological: Rotavirus; Biological: Pneumococcal 7-valent Conjugate Vaccine; Biological: HAV; Biological: MMR-V; Biological: DTaP
- LA4 (Infant Vaccines Only) (Experimental): Received vaccines:
  MenACWY: 12 and 15 months
  DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines: 2, 4, and 6 months
  DTaP, Hib: 15 months
  Pneumococcal, HAV, and MMR-V: 12 months
  Interventions: Biological: Meningococcal ACWY Conjugate Vaccine; Biological: DTaP-IPV-HBV; Biological: Hib; Biological: Rotavirus; Biological: Pneumococcal 7-valent Conjugate Vaccine; Biological: HAV; Biological: MMR-V; Biological: DTaP
- LA5 (MenACWY-CRM + Infant Vaccines) (Experimental): Received vaccines:
  MenACWY: 2, 4, 6, and 12 months
  DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines: 2, 4, and 6 months
  Pneumococcal, HAV, and MMR-V: 12 months
  Interventions: Biological: Meningococcal ACWY Conjugate Vaccine; Biological: DTaP-IPV-HBV; Biological: Hib; Biological: Rotavirus; Biological: Pneumococcal 7-valent Conjugate Vaccine; Biological: HAV; Biological: MMR-V
- LA6A (Infant Vaccines Only) (Experimental): Received vaccines:
  MenACWY: 12, and 15 months
  DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines: 2, 4, and 6 months
  Pneumococcal, HAV, and MMR-V: 12 months
  Interventions: Biological: Meningococcal ACWY Conjugate Vaccine; Biological: DTaP-IPV-HBV; Biological: Hib; Biological: Rotavirus; Biological: Pneumococcal 7-valent Conjugate Vaccine; Biological: HAV; Biological: MMR-V
- LA6B (Infant Vaccines Only) (Experimental): Received vaccines:
  MenACWY: 13 and 15 months
  DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines: 2, 4, and 6 months
  Pneumococcal, HAV, and MMR-V: 12 months
  Interventions: Biological: Meningococcal ACWY Conjugate Vaccine; Biological: DTaP-IPV-HBV; Biological: Hib; Biological: Rotavirus; Biological: Pneumococcal 7-valent Conjugate Vaccine; Biological: HAV; Biological: MMR-V
- LA6C (Infant Vaccines Only) (Experimental): Received vaccines:
  MenACWY: 18 months
  DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines: 2, 4, and 6 months
  Pneumococcal, HAV, and MMR-V: 12 months
  Interventions: Biological: Meningococcal ACWY Conjugate Vaccine; Biological: DTaP-IPV-HBV; Biological: Hib; Biological: Rotavirus; Biological: Pneumococcal 7-valent Conjugate Vaccine; Biological: HAV

INTERVENTIONS:
Biological: Meningococcal ACWY Conjugate Vaccine
  Other Names: Menveo
Biological: DTaP-IPV-HBV
  Other Names: Pediarix® (Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Hepatitis B (Recombinant) and Inactivated Poliovirus Vaccine Combined
Biological: Hib
  Other Names: ActHIB® (Haemophilus influenzae type b Conjugate Vaccine)
Biological: Rotavirus
  Other Names: RotaTeq® Rotavirus Vaccine, Live, Oral, Pentavalent
Biological: Pneumococcal 7-valent Conjugate Vaccine
  Other Names: Prevnar®
  Arms: LA1A (MenACWY-CRM + Infant Vaccines); LA1B (MenACWY-CRM + Infant Vaccines); LA2 (Infant Vaccines Only); LA3A (MenACWY-CRM + Infant Vaccines); LA3B (MenACWY-CRM + Infant Vaccines); LA4 (Infant Vaccines Only); LA5 (MenACWY-CRM + Infant Vaccines); LA6A (Infant Vaccines Only); LA6B (Infant Vaccines Only); LA6C (Infant Vaccines Only); US1A (MenACWY-CRM + Infant Vaccines); US1B (MenACWY-CRM + Infant Vaccines); US2 (Infant Vaccines Only); US3 (MenACWY-CRM + Infant Vaccines); US4B (Infant Vaccines Only); US4C (Infant Vaccines Only)
Biological: HAV
  Other Names: Havrix® (Hepatitis A Vaccine, Inactivated)
Biological: MMR-V
  Other Names: ProQuad™ (Measles, Mumps, Rubella and Varicella vaccine)
  Arms: LA1A (MenACWY-CRM + Infant Vaccines); LA1B (MenACWY-CRM + Infant Vaccines); LA2 (Infant Vaccines Only); LA3A (MenACWY-CRM + Infant Vaccines); LA3B (MenACWY-CRM + Infant Vaccines); LA4 (Infant Vaccines Only); LA5 (MenACWY-CRM + Infant Vaccines); LA6A (Infant Vaccines Only); LA6B (Infant Vaccines Only); US1A (MenACWY-CRM + Infant Vaccines); US1B (MenACWY-CRM + Infant Vaccines); US2 (Infant Vaccines Only); US3 (MenACWY-CRM + Infant Vaccines); US4A (Infant Vaccines Only); US4B (Infant Vaccines Only); US4C (Infant Vaccines Only)
Biological: DTaP
  Other Names: Infanrix® (Diphtheria and Tetanus Toxoids and Acellular Pertussis Vaccine Adsorbed)
  Arms: LA3A (MenACWY-CRM + Infant Vaccines); LA3B (MenACWY-CRM + Infant Vaccines); LA4 (Infant Vaccines Only)

SUMMARY:
This study will evaluate the safety and immune response of the Novartis Meningococcal ACWY conjugate vaccine when administered with routine infant vaccinations to healthy infants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term 2-month-old infants for whom a parent/legal representative has given written informed consent.

Exclusion Criteria:

* Subjects with a previous or suspected disease caused by Neisseria meningitidis, Corynebacterium diphtheriae, Clostridium tetani, Poliovirus, Hepatitis B, Haemophilus influenzae type b (Hib), Pneumococcus or Bordetella pertussis; previous immunization with a meningococcal vaccine or vaccine containing meningococcal antigen(s) or prior vaccination with Diptheria, Tetanus, Pertussis (acellular or whole cell), inactivated polio vaccineIPV or oral polio vaccineOPV, H. influenzae type b (Hib) or Pneumococcus; who have had household contact with and/or intimate exposure to an individual with laboratory confirmed N. meningitidis (serogroups A, C, W-135, or Y), B. pertussis, Hib, C. diphtheriae, Polio, or pneumococcal infection at any time since birth; Any serious acute, chronic or progressive disease

Ages: 2 Months to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4545 (Actual)
Dates: Start 2007-03; Primary Completion 2008-09 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis - Vaccines, Study Chair — Novartis Vaccines & Diagnostics
Locations (63):
- United States (53):
  - Growing Up Pediatrics, Bessemer, Alabama
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Growing Up Pediatrics, Birmingham, Alabama
  - Premier Health Research Center, LLC, Downey, California
  - Kaiser Permanente Oakland, Oakland, California
  - Kaiser Permanente Med Group - Vaccine Study Ctr, Oakland, California
  - Center for Clinical Trials, LLC, Paramount, California
  - Kaiser Permanente Pleasanton, Pleasanton, California
  - Kaiser Permanente Richmond, Richmond, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - Kaiser Permanente Santa Clara, Santa Clara, California
  - UCLA Center for Vaccine Research, Torrence, California
  - The Children's Hospital, Aurora, Colorado
  - Longmont Medical Research Network, Longmont, Colorado
  - Children's Memorial Hospital, Chicago, Illinois
  - Kentucky Pediatric/Adult Research Inc., Bardstown, Kentucky
  - Annapolis Pediatrics, Annapolis, Maryland
  - Center for Vaccine Development, Baltimore, Maryland
  - The Pediatric Center, Frederick, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - Pediatric Associates of Fall River, Fall River, Massachusetts
  - Creighton University, Omaha, Nebraska
  - Children's Physicians Dundee, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Montefiore Medical Center, The Bronx, New York
  - Akron Children's Hospital, Akron, Ohio
  - Louis P. Brine, Jr., MD, Beeghley Medical Park, Boardman, Ohio
  - Senders Pediatric Research at Dr. Senders and Associates, Cleveland, Ohio
  - Carnegie Pediatrics, Carnegie, Pennsylvania
  - Children's Health Care - West, Erie, Pennsylvania
  - UPMC/Community Medicine, Inc., Greenville, Pennsylvania
  - Family Healthcare Partners, Grove City, Pennsylvania
  - Pennridge Pediatric Associates, Harleyville, Pennsylvania
  - Pediatric Associates of Latrobe, Latrobe, Pennsylvania
  - Pediatric Medical Associates, Norristown, Pennsylvania
  - Squirrel Hill Office, Pittsburgh, Pennsylvania
  - Pediatric Alliance, Greentree Division, Pittsburgh, Pennsylvania
  - South Hills Pediatrics, Pittsburgh, Pennsylvania
  - Pediatric Alliance, Southwestern, Pittsburgh, Pennsylvania
  - Primary Physicians Research, Inc, Pittsburgh, Pennsylvania
  - Pediatrics Medical Associates, Rydal, Pennsylvania
  - Pennridge Pediatric Associates, Sellersville, Pennsylvania
  - Laurel Pediatrics, Uniontown, Pennsylvania
  - CCP - Pittsburgh Pediatrics, Wexford, Pennsylvania
  - Goodlettsville Pediatrics, Madison, Tennessee
  - Research Across America, Dallas, Texas
  - Mercury Pharma Services, Houston, Texas
  - Scott and White Hospital, Temple, Texas
  - Wee Care Pediatrics, Layton, Utah
  - Utah Valley Pediatrics - Timpanogos, Orem, Utah
  - Foothill Family Clinic, Salt Lake City, Utah
  - Copperview Medical Center, South Jordan, Utah
  - Monroe Medical Foundation, Monroe, Wisconsin
- Argentina (6):
  - CEDEPAP Rio IV, Alvear 1439 PB Dpto, Rio IV, Cordoba, Córdoba Province
  - Hospitales Materno Neonatal,, Castro Barros 650 - Barrio San Martin, Cordoba, Córdoba Province
  - CdePAP, Centro De Desarrollo De Proyectos Avanzados Roma 1465,, Córdoba, Córdoba Province
  - Hospital Regional Luis Pasteur,, Mendoza N°2152, Villa Maria, Cordoba,, Córdoba Province
  - Buenos Aires, Argentina, Buenos Aires
  - Centro Estudios Infect, Scalabrini Ortiz 676, Buenos Aires, Buenos Aires,
- Colombia (4):
  - Siloe, Calle 1 #50-51, Cali
  - Comfenalco, Calle 6#5-42, Cali
  - Hospital C H Trujillo, Calle 72U 28 F-00, Cali
  - Corporation Cientifica, Ped Calle 5B5 No.37 Bis-28, Cali

REFERENCES:
- [Result] Klein NP, Reisinger KS, Johnston W, Odrljin T, Gill CJ, Bedell L, Dull P. Safety and immunogenicity of a novel quadrivalent meningococcal CRM-conjugate vaccine given concomitantly with routine vaccinations in infants. Pediatr Infect Dis J. 2012 Jan;31(1):64-71. doi: 10.1097/INF.0b013e31823dce5c. PMID 22094635

RESULTS

PARTICIPANT FLOW:
Groups:
- US1A (MenACWY-CRM + Infant Vaccines): US infants received MenACWY at 2, 4 and 6 months of age along with routine infant vaccines, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccine. These infants received a fourth dose of MenACWY concomitantly with pneumococcal, HAV, and MMR-V vaccines at 12 months of age.
- US1B (MenACWY-CRM + Infant Vaccines): US infants received MenACWY at 2, 4 and 6 months of age along with routine infant vaccines, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines. These infants received pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and a fourth dose of MenACWY at 13 months of age.
- US2 (Infant Vaccines Only); US4A (Infant Vaccines Only): US infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. These infants received one dose of MenACWY concomitantly with pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and a second dose of MenACWY at 15 months of age.
- US3 (MenACWY-CRM + Infant Vaccines): US infants received MenACWY at 2, 4 and 6 months of age along with routine infant vaccines, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccine. These infants received fourth dose of MenACWY concomitantly with pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months of age.
- US4B (Infant Vaccines Only): US infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. These subjects received concomitant pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and one dose of MenACWY at 13 and a second dose of MenACWY at 15 months of age.
- US4C (Infant Vaccines Only): US infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines, at 2, 4 and 6 months of age. These subjects received concomitant pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months and one dose of MenACWY at 18 months of age.
- LA1A (MenACWY-CRM + Infant Vaccines): LA infants received MenACWY at 2 and 6 months of age; and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. These subjects received a third dose of MenACWY concomitantly with pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months of age.
- LA1B (MenACWY-CRM + Infant Vaccines): LA infants received MenACWY at 2 and 6 months of age and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. These subjects received pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months and a third dose of MenACWY at 13 months of age.
- LA2 (Infant Vaccines Only): LA infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. These infants received one dose of MenACWY concomitantly with pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and a second dose of MenACWY at 15 months of age.
- LA3A (MenACWY-CRM + Infant Vaccines): LA infants received MenACWY at 2, 4 and 6 months of age; and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, pneumococcal conjugate vaccine, and rotavirus vaccine. Around 12 months of age, these infants were recommended to receive pneumococcal conjugate vaccine, HAV, and MMR-V. At 16 months of age, these subjects received the fourth dose of MenACWY along with concomitant DTaP and Hib.
- LA3B (MenACWY-CRM + Infant Vaccines): LA infants received MenACWY at 2, 4 and 6 months of age; and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, pneumococcal conjugate vaccine, and rotavirus vaccine. Around 12 months of age, received pneumococcal conjugate vaccine, HAV, and MMR-V. At 16 months of age, these subjects received DTaP and Hib. At 17 months of age, these subjects received the fourth dose of MenACWY.
- LA4 (Infant Vaccines Only): LA infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, pneumococcal conjugate vaccine, and rotavirus vaccine at 2, 4 and 6 months of age. These infants received one dose of MenACWY concomitantly with pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months and a second dose of MenACWY along with DTaP and Hib vaccines at 15 months of age.
- LA5 (MenACWY-CRM + Infant Vaccines): LA infants received MenACWY at 2, 4 and 6 months of age; and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines. At 12 months of age, these subjects received the fourth dose of MenACWY concomitantly with pneumococcal conjugate vaccine, HAV, and MMR-V.
- LA6A (Infant Vaccines Only): LA infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus, and pneumococcal conjugate vaccines, at 2, 4 and 6 months of age. These infants received concomitant pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and one dose of MenACWY at 12 and a second dose of MenACWY at 15 months of age.
- LA6B (Infant Vaccines Only): LA infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus, and pneumococcal conjugate vaccines, at 2, 4 and 6 months of age. These infants received concomitant pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and one dose of MenACWY at 13 and a second dose of MenACWY at 15 months of age.
- LA6C (Infant Vaccines Only): LA infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus, and pneumococcal conjugate vaccines, at 2, 4 and 6 months of age. These infants received concomitant pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and one dose of MenACWY at 18 months of age
Period: Overall Study
Arm/Group | US1A (MenACWY-CRM + Infant Vaccines) | US1B (MenACWY-CRM + Infant Vaccines) | US2 (Infant Vaccines Only) | US3 (MenACWY-CRM + Infant Vaccines) | US4A (Infant Vaccines Only) | US4B (Infant Vaccines Only) | US4C (Infant Vaccines Only) | LA1A (MenACWY-CRM + Infant Vaccines) | LA1B (MenACWY-CRM + Infant Vaccines) | LA2 (Infant Vaccines Only) | LA3A (MenACWY-CRM + Infant Vaccines) | LA3B (MenACWY-CRM + Infant Vaccines) | LA4 (Infant Vaccines Only) | LA5 (MenACWY-CRM + Infant Vaccines) | LA6A (Infant Vaccines Only) | LA6B (Infant Vaccines Only) | LA6C (Infant Vaccines Only)
Started | 154 | 166 | 159 | 680 | 76 | 70 | 203 | 151 | 150 | 148 | 151 | 150 | 150 | 1426 | 358 | 170 | 183
Completed | 121 | 120 | 110 | 561 | 8 | 54 | 178 | 145 | 144 | 121 | 141 | 139 | 135 | 1270 | 281 | 152 | 174
Not Completed | 33 | 46 | 49 | 119 | 68 | 16 | 25 | 6 | 6 | 27 | 10 | 11 | 15 | 156 | 77 | 18 | 9
Not completed — ADMINISTRATIVE REASON | 11 | 9 | 9 | 20 | 9 | 1 | 1 | 0 | 2 | 1 | 1 | 1 | 1 | 1 | 2 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 2 | 4 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Not completed — INAPPROPRIATE ENROLLMENT | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Not completed — Lost to Follow-up | 8 | 6 | 13 | 29 | 11 | 5 | 8 | 1 | 0 | 6 | 2 | 4 | 6 | 74 | 29 | 4 | 5
Not completed — Protocol Violation | 2 | 6 | 4 | 12 | 3 | 1 | 3 | 0 | 0 | 4 | 2 | 2 | 4 | 19 | 9 | 6 | 2
Not completed — UNABLE TO CLASSIFY | 1 | 0 | 0 | 1 | 3 | 2 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 20 | 12 | 6 | 1
Not completed — Withdrawal by Subject | 9 | 24 | 21 | 52 | 38 | 6 | 12 | 4 | 4 | 13 | 5 | 4 | 4 | 37 | 22 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- TOTAL: Total of all reporting groups
Arm/Group | US1A (MenACWY-CRM + Infant Vaccines) | US1B (MenACWY-CRM + Infant Vaccines) | US2 (Infant Vaccines Only) | US3 (MenACWY-CRM + Infant Vaccines) | US4A (Infant Vaccines Only) | US4B (Infant Vaccines Only) | US4C (Infant Vaccines Only) | LA1A (MenACWY-CRM + Infant Vaccines) | LA1B (MenACWY-CRM + Infant Vaccines) | LA2 (Infant Vaccines Only) | LA3A (MenACWY-CRM + Infant Vaccines) | LA3B (MenACWY-CRM + Infant Vaccines) | LA4 (Infant Vaccines Only) | LA5 (MenACWY-CRM + Infant Vaccines) | LA6A (Infant Vaccines Only) | LA6B (Infant Vaccines Only) | LA6C (Infant Vaccines Only) | TOTAL
Number analyzed (Participants) | 154 | 166 | 159 | 680 | 76 | 70 | 203 | 151 | 150 | 148 | 151 | 150 | 150 | 1426 | 358 | 170 | 183 | 4545
Age, Continuous [Mean (Standard Deviation); unit: days] | 66.1 (7.2) | 65.8 (6.6) | 65.7 (6.5) | 65.0 (6.0) | 66.1 (6.2) | 65.0 (6.5) | 65.9 (6.5) | 68.0 (7.7) | 68.6 (8.9) | 67.8 (8.3) | 67.0 (7.9) | 68.4 (8.7) | 67.5 (8.0) | 65.0 (9.4) | 67.7 (9.7) | 59.5 (6.2) | 65.0 (7.9) | 65.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 72 | 71 | 340 | 39 | 29 | 103 | 79 | 82 | 72 | 72 | 75 | 81 | 682 | 178 | 89 | 91 | 2223
  Male | 86 | 94 | 88 | 340 | 37 | 41 | 100 | 72 | 68 | 76 | 79 | 75 | 69 | 744 | 180 | 81 | 92 | 2322

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With hSBA Titer >=1:8 - US Subjects
Description: Immunogenicity as measured by percentage of subjects with hSBA titer >=1:8 directed against N. meningitidis serogroups A, C, W and Y; after four doses of MenACWY-CRM at 2, 4, and 6 and 12 months of age
Time Frame: 13 months of age (one month post-toddler vaccination)
Population: The analysis was done on per protocol population
  Per protocol was defined as subjects who:
  * received all the relevant doses of vaccine correctly
  * provided evaluable serum samples at the relevant time points
  * had no major protocol deviation as defined prior to database lock
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- US1A (MenACWY- CRM + Infant Vaccines): US infants received one dose of MenACWY at 2, 4 and 6 months of age and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, pneumococcal conjugate vaccine, and rotavirus vaccine.At 12 months of age received fourth dose of MenACWY along with concomitant pneumococcal,HAV, and MMR-V vaccines.
- US2 (Infant Vaccine Only): received as part of routine infant vaccination schedule DTaP-IPV-HBV,Hib, pneumococcal conjugate vaccine, and rotavirus vaccine at 2, 4 and 6 months of age. At 12 months of age, these subjects received a dose of MenACWY along with concomitant pneumococcal conjugate vaccine, HAV, and MMR-V. At 15 months of age, these subjects received a second dose of MenACWY.
Arm/Group | US1A (MenACWY- CRM + Infant Vaccines) | US2 (Infant Vaccine Only)
Number analyzed (Participants) | 86 | 74
Percentages of subjects
  A (84, 74) | 94 [87 to 98] | 72 [60 to 81]
  C (86, 73) | 98 [92 to 100] | 90 [81 to 96]
  W (85, 73) | 100 [96 to 100] | 58 [45 to 69]
  Y (84, 68) | 100 [96 to 100] | 56 [43 to 68]

2. Secondary Outcome: Number of Subjects With Solicited Local and Systemic Reactions Post First Vaccination - Infant Series
Description: Solicited local and systemic reactions post first vaccination of infant series were compared in subjects receiving Infant Vaccines only and subjects receiving MenACWY-CRM concomitantly with Infant Vaccines.
Time Frame: 7 days after vaccination
Population: The population used in analysis was the safety set Safety population was defined as: all subjects in the exposed population who provided post-baseline safety data. If a subject received an entirely wrong vaccine schedule (e.g., US3 instead of US4), the subject would be analyzed for safety according to the group the subject actually followed.
Measure: Number; unit: Subjects
Groups:
- US1B (MenACWY-CRM + Infant Vaccines ): US infants received MenACWY at 2, 4 and 6 months of age along with routine infant vaccines, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines. These infants received pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and a fourth dose of MenACWY at 13 months of age.
- US1 (MenACWY-CRM + Infant Vaccines): US infants received one dose of MenACWY at 2, 4 and 6 months of age; and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines. Group US1 was randomized into US1A and US1B subgroups.
- US4 (Infant Vaccines Only ): US infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. These infants received concomitant pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months of age. These infants were randomized in subgroup US4A, US4B and US4C.
- LA1 (MenACWY-CRM + Infant Vaccines): LA infants received MenACWY at 2 and 6 months of age and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. Group LA1 was randomized into LA1A and LA 1B subgroups.
- LA3 (MenACWY-CRM + Infant Vaccines): LA infants received MenACWY at 2, 4 and 6 months of age; and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, pneumococcal conjugate vaccine, and rotavirus vaccine. Group LA3 was further randomized into LA3A and LA3B subgroups.
- LA6 (Infant Vaccines Only): LA infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus, and pneumococcal conjugate vaccines, at 2, 4 and 6 months of age. These infants received concomitant pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months of age. Group LA6 was further randomized into LA6A and LA6B and LA6C subgroups.
Arm/Group | US1A (MenACWY-CRM + Infant Vaccines) | US1B (MenACWY-CRM + Infant Vaccines ) | US1 (MenACWY-CRM + Infant Vaccines) | US2 (Infant Vaccines Only) | US3 (MenACWY-CRM + Infant Vaccines) | US4 (Infant Vaccines Only ) | LA1 (MenACWY-CRM + Infant Vaccines) | LA2 (Infant Vaccines Only) | LA3 (MenACWY-CRM + Infant Vaccines) | LA4 (Infant Vaccines Only) | LA5 (MenACWY-CRM + Infant Vaccines) | LA6 (Infant Vaccines Only)
Number analyzed (Participants) | 153 | 165 | 318 | 159 | 677 | 345 | 301 | 148 | 301 | 150 | 1424 | 709
Subjects
  Erythema (mm) - Any | 10 | 17 | 27 | 23 | 66 | 54 | 86 | 62 | 86 | 65 | 542 | 273
  Erythema (mm) - Severe | 0 | 0 | 0 | 2 | 0 | 4 | 0 | 0 | 1 | 1 | 1 | 4
  Induration (mm) - Any | 10 | 14 | 24 | 25 | 61 | 44 | 74 | 56 | 72 | 53 | 249 | 126
  Induration (mm) - Severe | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0
  Tenderness - Any | 64 | 76 | 140 | 69 | 324 | 161 | 154 | 96 | 170 | 95 | 916 | 501
  Tenderness - Severe | 3 | 4 | 7 | 6 | 25 | 19 | 30 | 19 | 22 | 20 | 92 | 74
  Body Temp. ( >= 38° C ) | 13 | 6 | 19 | 7 | 32 | 21 | 15 | 12 | 18 | 5 | 211 | 97
  Change in Eating Habits - Any | 42 | 46 | 88 | 34 | 171 | 96 | 37 | 30 | 44 | 16 | 250 | 127
  Change in Eating Habits - Severe | 1 | 1 | 2 | 1 | 8 | 2 | 2 | 0 | 0 | 1 | 6 | 4
  Diarrhea - Any | 24 | 23 | 47 | 17 | 107 | 46 | 42 | 20 | 44 | 22 | 222 | 96
  Diarrhea - Severe | 2 | 0 | 2 | 1 | 3 | 1 | 1 | 0 | 1 | 0 | 2 | 2
  Irritability - Any | 82 | 107 | 189 | 96 | 419 | 211 | 121 | 62 | 99 | 59 | 508 | 240
  Irritability - Severe | 6 | 2 | 8 | 4 | 24 | 12 | 7 | 2 | 4 | 2 | 22 | 2
  Persistent Crying - Any | 43 | 74 | 117 | 49 | 252 | 125 | 95 | 53 | 87 | 43 | 479 | 258
  Persistent Crying - Severe | 1 | 2 | 3 | 5 | 11 | 8 | 5 | 3 | 11 | 8 | 29 | 21
  Rash - Any | 6 | 9 | 15 | 5 | 16 | 11 | 11 | 6 | 12 | 4 | 98 | 55
  Rash - Severe | 3 | 4 | 7 | 3 | 4 | 3 | 7 | 2 | 4 | 1 | 54 | 26
  Sleepiness - Any | 83 | 104 | 187 | 76 | 354 | 173 | 106 | 53 | 93 | 52 | 727 | 381
  Sleepiness - Severe | 2 | 3 | 5 | 0 | 14 | 3 | 8 | 2 | 6 | 4 | 21 | 14
  Vomiting - Any | 15 | 18 | 33 | 14 | 67 | 36 | 25 | 9 | 29 | 17 | 215 | 100
  Vomiting - Severe | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 1
  Analgesic / Antipyretic medication used | 105 | 120 | 225 | 110 | 447 | 223 | 155 | 75 | 159 | 80 | 996 | 510

3. Secondary Outcome: Number of Subjects With Solicited Local and Systemic Reactions Post Second Vaccination - Infant Series
Description: Solicited local and systemic reactions post second vaccination of infant series were compared in subjects receiving Infant Vaccines only and subjects receiving MenACWY-CRM concomitantly with Infant Vaccines.
Time Frame: 7 days after vaccination
Population: The population used in analysis was the safety set: The total number of subjects analyzed was less than the safety set due to subject withdrawals. LA1 and LA 2 groups are not included here as they did not receive MenACWY at 4 months of age.
Measure: Number; unit: Subjects
Groups:
- US4 (Infant Vaccines Only): US infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. These infants received concomitant pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months of age. These infants were randomized in subgroup US4A, US4B and US4C.
Arm/Group | US1A (MenACWY-CRM + Infant Vaccines) | US1B (MenACWY-CRM + Infant Vaccines) | US1 (MenACWY-CRM + Infant Vaccines) | US2 (Infant Vaccines Only) | US3 (MenACWY-CRM + Infant Vaccines) | US4 (Infant Vaccines Only) | LA3 (MenACWY-CRM + Infant Vaccines) | LA4 (Infant Vaccines Only) | LA5 (MenACWY-CRM + Infant Vaccines) | LA6 (Infant Vaccines Only)
Number analyzed (Participants) | 141 | 150 | 291 | 151 | 645 | 325 | 301 | 150 | 1424 | 709
Subjects
  Erythema (mm) - Any | 14 | 19 | 33 | 35 | 75 | 60 | 92 | 45 | 583 | 311
  Erythema (mm) - Severe | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Induration (mm) - Any | 16 | 16 | 32 | 27 | 45 | 48 | 73 | 36 | 194 | 126
  Induration (mm) - Severe | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0
  Tenderness - Any | 59 | 59 | 118 | 56 | 230 | 137 | 115 | 59 | 726 | 401
  Tenderness - Severe | 1 | 0 | 1 | 2 | 13 | 11 | 13 | 5 | 49 | 45
  Body Temp. ( >= 38° C ) | 17 | 6 | 23 | 15 | 49 | 28 | 23 | 13 | 223 | 122
  Change in Eating Habits - Any | 25 | 21 | 46 | 20 | 122 | 64 | 28 | 12 | 160 | 90
  Change in Eating Habits - Severe | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 0 | 6 | 5
  Diarrhea - Any | 16 | 10 | 26 | 11 | 53 | 35 | 28 | 14 | 149 | 90
  Diarrhea - Severe | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 4 | 1
  Irritability - Any | 83 | 80 | 163 | 83 | 342 | 182 | 82 | 41 | 414 | 209
  Irritability - Severe | 2 | 0 | 2 | 3 | 14 | 9 | 3 | 0 | 13 | 5
  Persistent Crying - Any | 42 | 41 | 83 | 34 | 178 | 107 | 42 | 22 | 294 | 187
  Persistent Crying - Severe | 0 | 0 | 0 | 0 | 5 | 4 | 4 | 1 | 14 | 10
  Rash - Any | 3 | 5 | 8 | 4 | 24 | 13 | 13 | 2 | 97 | 46
  Rash - Severe | 3 | 1 | 4 | 1 | 6 | 4 | 5 | 1 | 52 | 29
  Sleepiness - Any | 69 | 56 | 125 | 47 | 238 | 131 | 62 | 26 | 485 | 237
  Sleepiness - Severe | 0 | 0 | 0 | 1 | 3 | 2 | 4 | 1 | 13 | 7
  Vomiting - Any | 8 | 9 | 17 | 7 | 49 | 27 | 20 | 10 | 136 | 75
  Vomiting - Severe | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0
  Analgesic / Antipyretic medication used | 94 | 91 | 185 | 96 | 385 | 201 | 131 | 61 | 857 | 430

4. Primary Outcome: Geometric Mean hSBA Titers - US Subjects
Description: Immunogenicity as measured by Geometric Mean hSBA Titers directed against N. meningitidis serogroups A, C, W and Y; comparison of four doses of MenACWY-CRM at 2, 4, and 6 and 12 months of age versus a single dose at 12 months of age.
Time Frame: 13 months of age (one month post-toddler vaccination)
Population: The analysis was done on per protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- US1A (MenACWY- CRM + Infant Vaccines ): US infants received one dose of MenACWY at 2, 4 and 6 months of age and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, pneumococcal conjugate vaccine, and rotavirus vaccine.At 12 months of age received fourth dose of MenACWY along with concomitant pneumococcal,HAV, and MMR-V vaccines.
Arm/Group | US1A (MenACWY- CRM + Infant Vaccines ) | US2 (Infant Vaccine Only)
Number analyzed (Participants) | 86 | 74
Titers
  A Pre-vaccination (84, 74) | 2.51 [2.14 to 2.96] | 2.14 [1.8 to 2.54]
  A Post-vaccination (84, 74) | 77 [55 to 109] | 17 [12 to 25]
  C Pre-vaccination (86, 73) | 7.72 [5.9 to 10] | 2.26 [1.69 to 3.03]
  C Post-vaccination (86, 73) | 227 [155 to 332] | 35 [23 to 54]
  W Pre-vaccination (85, 73) | 14 [11 to 18] | 2.21 [1.69 to 2.9]
  W Post-vaccination (85, 73) | 416 [288 to 602] | 11 [7.59 to 17]
  Y Pre-vaccination (84, 68) | 11 [8.76 to 15] | 2.14 [1.6 to 2.86]
  Y Post-vaccination (84, 68) | 395 [269 to 580] | 10 [6.72 to 16]
Statistical Analysis 1: Comparison: US1A (MenACWY- CRM + Infant Vaccines ) vs US2 (Infant Vaccine Only); Using the MenACWY GMTs, immunogenicity of the fourth dose at 1 month after the 12-month vaccination in those subjects receiving MenACWY at 2, 4, and 6 months was considered superior to the immune response of a single dose given at 12-months of age if the lower limit of the two-sided 95% CI of the ratio of the two GMTs was >= 2.0; Test type: Superiority or Other; ANOVA; Ratio of GMTs = 4.53, 95% CI 2-sided [3.04 to 6.74] — A (Post-vaccination GMT; group ratio US1A:US2)
Statistical Analysis 2: Comparison: US1A (MenACWY- CRM + Infant Vaccines ) vs US2 (Infant Vaccine Only); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; ANOVA; Ratio of GMTs = 6.39, 95% CI 2-sided [4.16 to 9.79] — C (Post-vaccination GMT; group ratio US1A:US2)
Statistical Analysis 3: Comparison: US1A (MenACWY- CRM + Infant Vaccines ) vs US2 (Infant Vaccine Only); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; ANOVA; Ratio of GMTs = 37, 95% CI 2-sided [24 to 58] — W (Post-vaccination GMT; group ratio US1A:US2)
Statistical Analysis 4: Comparison: US1A (MenACWY- CRM + Infant Vaccines ) vs US2 (Infant Vaccine Only); Using the MenACWY GMTs, immunogenicity of the fourth dose at 1 month after the 12-month vaccination in those subjects receiving MenACWY at 2, 4, and 6 months was considered superior to the immune response of a single dose given at 12-months of age if the lower limit of the two-sided 95% CI of the ratio of the two GMTs was >= 2.0. Ratio of GMTs; Test type: Superiority or Other; ANOVA; Ratio of GMTs = 38, 95% CI 2-sided [24 to 60] — Y (Post-vaccination GMT; group ratio US1A:US2)

5. Secondary Outcome: Number of Subjects With Solicited Local and Systemic Reactions Post Third Vaccination - Infant Series
Description: Solicited local and systemic reactions post third vaccination of infant series were compared in subjects receiving Infant Vaccines only and subjects receiving MenACWY-CRM concomitantly with Infant Vaccines.
Time Frame: 7 days after vaccination
Population: The population used in analysis was the safety set: The total number of subjects analyzed was less than the safety set due to subject withdrawals.
Measure: Number; unit: Subjects
Arm/Group | US1A (MenACWY-CRM + Infant Vaccines) | US1B (MenACWY-CRM + Infant Vaccines) | US1 (MenACWY-CRM + Infant Vaccines) | US2 (Infant Vaccines Only) | US3 (MenACWY-CRM + Infant Vaccines) | US4 (Infant Vaccines Only) | LA1 (MenACWY-CRM + Infant Vaccines) | LA2 (Infant Vaccines Only) | LA3 (MenACWY-CRM + Infant Vaccines) | LA4 (Infant Vaccines Only) | LA5 (MenACWY-CRM + Infant Vaccines) | LA6 (Infant Vaccines Only)
Number analyzed (Participants) | 138 | 145 | 283 | 143 | 627 | 311 | 297 | 131 | 290 | 147 | 1357 | 679
Subjects
  Erythema (mm) - Any | 16 | 18 | 34 | 28 | 92 | 67 | 69 | 27 | 64 | 38 | 485 | 273
  Erythema (mm) - Severe | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
  Induration (mm) - Any | 15 | 15 | 30 | 29 | 59 | 53 | 54 | 25 | 64 | 32 | 125 | 73
  Induration (mm) - Severe | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Tenderness - Any | 37 | 45 | 82 | 45 | 189 | 92 | 92 | 40 | 78 | 50 | 504 | 306
  Tenderness - Severe | 0 | 0 | 0 | 1 | 1 | 7 | 6 | 2 | 2 | 1 | 21 | 14
  Body Temp. ( >= 38° C ) | 4 | 9 | 13 | 14 | 33 | 20 | 13 | 10 | 26 | 14 | 164 | 101
  Change in Eating Habits - Any | 19 | 22 | 41 | 18 | 94 | 39 | 25 | 11 | 23 | 9 | 126 | 66
  Change in Eating Habits - Severe | 0 | 0 | 0 | 1 | 3 | 2 | 1 | 1 | 1 | 0 | 5 | 3
  Diarrhea - Any | 13 | 9 | 22 | 9 | 41 | 26 | 17 | 8 | 12 | 11 | 97 | 58
  Diarrhea - Severe | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 2 | 3
  Irritability - Any | 58 | 73 | 131 | 70 | 285 | 157 | 57 | 29 | 62 | 28 | 311 | 164
  Irritability - Severe | 1 | 1 | 2 | 0 | 4 | 6 | 0 | 1 | 2 | 0 | 5 | 2
  Persistent Crying - Any | 28 | 26 | 54 | 24 | 135 | 74 | 28 | 15 | 27 | 12 | 181 | 118
  Persistent Crying - Severe | 0 | 0 | 0 | 0 | 4 | 4 | 2 | 2 | 0 | 0 | 11 | 2
  Rash - Any | 2 | 9 | 11 | 4 | 14 | 8 | 8 | 1 | 6 | 1 | 62 | 29
  Rash - Severe | 1 | 4 | 5 | 3 | 2 | 1 | 5 | 0 | 3 | 1 | 29 | 10
  Sleepiness - Any | 37 | 41 | 78 | 39 | 179 | 91 | 38 | 15 | 45 | 17 | 317 | 164
  Sleepiness - Severe | 0 | 0 | 0 | 0 | 6 | 1 | 1 | 0 | 1 | 0 | 6 | 3
  Vomiting - Any | 6 | 6 | 12 | 9 | 31 | 20 | 16 | 9 | 11 | 12 | 104 | 52
  Vomiting - Severe | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 1
  Analgesic / Antipyretic medication used | 75 | 82 | 157 | 96 | 349 | 178 | 93 | 38 | 90 | 51 | 592 | 342

6. Secondary Outcome: Number of Subjects With Solicited Local and Systemic Reactions After Vaccination at 12 Months of Age
Description: Solicited local and systemic reactions after receiving MenACWY-CRM vaccination at 12 months of age were compared in subjects receiving Infant Vaccines only and subjects receiving MenACWY-CRM concomitantly with Infant Vaccines.
Time Frame: 7 days after vaccination
Population: as for outcome 5
Measure: Number; unit: Subjects
Groups:
- US1A + US3 (MenACWY-CRM + Infant Vaccines): Groups MenACWY-CRM + infant vaccines (US1A and US3) Pooled. In both groups US infants received MenACWY at 2, 4 and 6 months of age along with routine infant vaccines, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccine. These infants received a fourth dose of MenACWY concomitantly with pneumococcal, HAV, and MMR-V vaccines at 12 months of age.
- US2 + US4A (Infant Vaccines Only): Groups Infant Vaccines only (US2 and US4A) pooled.
  In both groups US infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. These infants received one dose of MenACWY concomitantly with pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and a second dose of MenACWY at 15 months of age.
- US4B + US4C (Infant Vaccines Only): Groups Infant Vaccines only (US4B and US4C) pooled.
  Infant Vaccines only (US4B): US infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. These subjects received concomitant pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and either received one dose of MenACWY at 13 and and a second dose of MenACWY at 15 months of age (US4B); or one dose at 18 months of age (US4C).
- LA2 + LA4 + LA6A (Infant Vaccines Only): Groups Infant Vaccines only (LA2, LA4 and LA6A) pooled. In all groups LA infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. These infants received one dose of MenACWY concomitantly with pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and a second dose of MenACWY at 15 months of age.
- LA6B + LA6C (Infant Vaccines Only): Groups Infant Vaccines only LA6B and LA6C pooled.
  Infant Vaccines only (LA6B): LA infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus, and pneumococcal conjugate vaccines, at 2, 4 and 6 months of age. These infants received concomitant pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and either one dose of MenACWY at 13 and a second dose of MenACWY at 15 months of age (LA6B) or one dose of MenACWY at 18 months of age (LA6C).
Arm/Group | US1A (MenACWY-CRM + Infant Vaccines) | US1B (MenACWY-CRM + Infant Vaccines) | US1A + US3 (MenACWY-CRM + Infant Vaccines) | US2 + US4A (Infant Vaccines Only) | US3 (MenACWY-CRM + Infant Vaccines) | US4B + US4C (Infant Vaccines Only) | LA1A (MenACWY-CRM + Infant Vaccines) | LA1B (MenACWY-CRM + Infant Vaccines) | LA2 + LA4 + LA6A (Infant Vaccines Only) | LA5 (MenACWY-CRM + Infant Vaccines) | LA6B + LA6C (Infant Vaccines Only)
Number analyzed (Participants) | 122 | 124 | 704 | 137 | 582 | 261 | 145 | 143 | 564 | 1275 | 349
Subjects
  Erythema (mm) - Any | 11 | 16 | 81 | 18 | 70 | 49 | 36 | 33 | 166 | 309 | 67
  Erythema (mm) - Severe | 0 | 0 | 2 | 1 | 2 | 1 | 0 | 1 | 2 | 0 | 0
  Induration (mm) - Any | 10 | 13 | 44 | 12 | 34 | 39 | 32 | 28 | 72 | 84 | 43
  Induration (mm) - Severe | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
  Tenderness - Any | 28 | 31 | 177 | 38 | 149 | 75 | 35 | 32 | 184 | 392 | 100
  Tenderness - Severe | 0 | 0 | 2 | 0 | 2 | 1 | 6 | 2 | 2 | 8 | 3
  Body Temp. ( >= 38° C ) | 14 | 10 | 49 | 12 | 35 | 20 | 16 | 12 | 84 | 188 | 40
  Change in Eating Habits - Any | 21 | 17 | 101 | 20 | 80 | 29 | 10 | 11 | 56 | 138 | 46
  Change in Eating Habits - Severe | 1 | 2 | 7 | 1 | 6 | 1 | 1 | 0 | 4 | 5 | 0
  Diarrhea - Any | 5 | 14 | 61 | 16 | 56 | 14 | 9 | 10 | 51 | 123 | 37
  Diarrhea - Severe | 0 | 0 | 4 | 1 | 4 | 1 | 0 | 0 | 5 | 7 | 1
  Irritability - Any | 53 | 53 | 271 | 62 | 218 | 103 | 29 | 23 | 130 | 289 | 74
  Irritability - Severe | 2 | 2 | 8 | 4 | 6 | 1 | 1 | 2 | 5 | 3 | 0
  Persistent Crying - Any | 21 | 21 | 120 | 24 | 99 | 55 | 7 | 12 | 52 | 134 | 28
  Persistent Crying - Severe | 0 | 0 | 6 | 1 | 6 | 1 | 0 | 1 | 0 | 2 | 0
  Rash - Any | 8 | 4 | 31 | 5 | 23 | 12 | 3 | 1 | 20 | 65 | 17
  Rash - Severe | 1 | 1 | 3 | 3 | 2 | 3 | 2 | 0 | 8 | 36 | 10
  Sleepiness - Any | 38 | 29 | 149 | 22 | 111 | 50 | 18 | 15 | 81 | 211 | 53
  Sleepiness - Severe | 0 | 1 | 3 | 1 | 3 | 3 | 0 | 0 | 1 | 3 | 2
  Vomiting - Any | 6 | 4 | 27 | 8 | 21 | 11 | 3 | 5 | 35 | 82 | 12
  Vomiting - Severe | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 4 | 0
  Analgesic / Antipyretic medication used | 60 | 56 | 320 | 78 | 260 | 120 | 48 | 43 | 204 | 406 | 87

7. Secondary Outcome: Number of Subjects With Solicited Local and Systemic Reactions Post First Vaccination - Toddler Series
Description: Solicited local and systemic reactions post first vaccination of toddler series were compared in subjects receiving Infant Vaccines only and subjects receiving MenACWY-CRM concomitantly with Infant Vaccines.
Time Frame: 7 days post vaccination
Population: as for outcome 5
Measure: Number; unit: Subjects
Groups:
- US1A + US3 (MenACWY-CRM + Infant Vaccines): Groups MenACWY-CRM + infant vaccines (US1A and US3) Pooled.In both groups US infants received MenACWY at 2, 4 and 6 months of age along with routine infant vaccines, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccine. These infants received a fourth dose of MenACWY concomitantly with pneumococcal, HAV, and MMR-V vaccines at 12 months of age.
- US4B (Infant Vaccines Only): US infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. These subjects received concomitant pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and one dose of MenACWY at 13 and one dose at 15 months of age.
- LA6B (Infant Vaccines Only): LA infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus, and pneumococcal conjugate vaccines, at 2, 4 and 6 months of age. These infants received concomitant pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and one dose of MenACWY at 13 and one dose at 15 months of age.
Arm/Group | US1B (MenACWY-CRM + Infant Vaccines) | US1A + US3 (MenACWY-CRM + Infant Vaccines) | US2 + US4A (Infant Vaccines Only) | US4B (Infant Vaccines Only) | US4C (Infant Vaccines Only) | LA1A (MenACWY-CRM + Infant Vaccines) | LA1B (MenACWY-CRM + Infant Vaccines) | LA2 + LA4 + LA6A (Infant Vaccines Only) | LA3A (MenACWY-CRM + Infant Vaccines) | LA3B (MenACWY-CRM + Infant Vaccines) | LA5 (MenACWY-CRM + Infant Vaccines) | LA6B (Infant Vaccines Only) | LA6C (Infant Vaccines Only)
Number analyzed (Participants) | 120 | 704 | 136 | 59 | 179 | 145 | 143 | 564 | 142 | 137 | 1275 | 160 | 175
Subjects
  Erythema (mm) - Any | 7 | 81 | 18 | 9 | 28 | 36 | 17 | 166 | 36 | 19 | 309 | 24 | 52
  Erythema (mm) - Severe | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 7
  Induration (mm) - Any | 1 | 44 | 12 | 3 | 14 | 32 | 9 | 72 | 33 | 16 | 84 | 5 | 35
  Induration (mm) - Severe | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 5
  Tenderness - Any | 16 | 177 | 38 | 10 | 38 | 35 | 21 | 184 | 36 | 18 | 392 | 34 | 45
  Tenderness - Severe | 0 | 2 | 0 | 1 | 1 | 6 | 1 | 2 | 2 | 2 | 8 | 0 | 5
  Body Temp. ( >= 38° C ) | 5 | 49 | 12 | 0 | 5 | 16 | 5 | 84 | 4 | 2 | 188 | 7 | 8
  Change in Eating Habits - Any | 9 | 101 | 20 | 5 | 14 | 10 | 4 | 56 | 6 | 6 | 138 | 9 | 17
  Change in Eating Habits - Severe | 0 | 7 | 1 | 0 | 1 | 1 | 1 | 4 | 1 | 0 | 5 | 0 | 0
  Diarrhea - Any | 8 | 61 | 16 | 5 | 13 | 9 | 4 | 51 | 8 | 2 | 123 | 6 | 12
  Diarrhea - Severe | 0 | 4 | 1 | 2 | 1 | 0 | 0 | 5 | 0 | 1 | 7 | 0 | 0
  Irritability - Any | 39 | 271 | 62 | 17 | 52 | 29 | 10 | 130 | 13 | 9 | 289 | 25 | 28
  Irritability - Severe | 1 | 8 | 4 | 1 | 1 | 1 | 0 | 5 | 0 | 0 | 3 | 1 | 0
  Persistent Crying - Any | 16 | 120 | 24 | 10 | 17 | 7 | 5 | 52 | 4 | 5 | 134 | 9 | 15
  Persistent Crying - Severe | 0 | 6 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
  Rash - Any | 1 | 31 | 5 | 2 | 5 | 3 | 1 | 20 | 2 | 1 | 65 | 2 | 2
  Rash - Severe | 0 | 3 | 3 | 0 | 2 | 2 | 1 | 8 | 2 | 0 | 36 | 0 | 1
  Sleepiness - Any | 25 | 149 | 22 | 6 | 21 | 18 | 3 | 81 | 6 | 7 | 211 | 14 | 20
  Sleepiness - Severe | 1 | 3 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 1
  Vomiting - Any | 2 | 27 | 8 | 2 | 6 | 3 | 0 | 35 | 1 | 3 | 82 | 4 | 3
  Vomiting - Severe | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 4 | 0 | 0
  Analgesic / Antipyretic medication used | 37 | 320 | 77 | 16 | 45 | 48 | 15 | 204 | 20 | 8 | 406 | 14 | 34

8. Secondary Outcome: Number of Subjects With Solicited Local and Systemic Reactions Post Second Vaccination - Toddler Series
Description: Solicited local and systemic reactions post second vaccination of toddler series at 15 months of age.
Time Frame: 7 days post vaccination
Population: The population used in analysis was the safety set: The total number of subjects analyzed was less than the safety set due to subject withdrawals. Only subjects who received the second dose at 15 months were included in this analysis.
Measure: Number; unit: Subjects
Arm/Group | US2 + US4A (Infant Vaccines Only) | US4B (Infant Vaccines Only) | LA2 + LA4 + LA6A (Infant Vaccines Only) | LA6B (Infant Vaccines Only)
Number analyzed (Participants) | 120 | 55 | 539 | 153
Subjects
  Erythema (mm) - Any | 14 | 6 | 143 | 28
  Erythema (mm) - Severe | 0 | 1 | 2 | 0
  Induration (mm) - Any | 10 | 2 | 51 | 2
  Induration (mm) - Severe | 0 | 1 | 1 | 0
  Tenderness - Any | 19 | 16 | 128 | 33
  Tenderness - Severe | 0 | 0 | 5 | 1
  Body Temp. ( >= 38° C ) | 5 | 1 | 30 | 15
  Change in Eating Habits - Any | 7 | 2 | 18 | 11
  Change in Eating Habits - Severe | 0 | 0 | 0 | 1
  Diarrhea - Any | 4 | 3 | 28 | 9
  Diarrhea - Severe | 1 | 0 | 1 | 0
  Irritability - Any | 31 | 22 | 71 | 32
  Irritability - Severe | 0 | 0 | 2 | 1
  Persistent Crying - Any | 9 | 10 | 37 | 6
  Persistent Crying - Severe | 0 | 0 | 3 | 2
  Rash - Any | 4 | 1 | 9 | 3
  Rash - Severe | 0 | 0 | 4 | 3
  Sleepiness - Any | 12 | 8 | 36 | 12
  Sleepiness - Severe | 0 | 0 | 1 | 2
  Vomiting - Any | 5 | 2 | 12 | 7
  Vomiting - Severe | 0 | 0 | 0 | 0
  Analgesic / Antipyretic medication used | 40 | 14 | 85 | 21

9. Secondary Outcome: Number of Subjects With Solicited Local and Systemic Reactions Post First Vaccination - Infant Series
Description: Solicited local and systemic reactions reported post first vaccination was compared in subjects receiving MenACWY versus Hib Vaccines.
Time Frame: 7 days post-vaccination
Population: as for outcome 5
Measure: Number; unit: Subjects
Groups:
- US1 + US3 (Men ACWY-CRM + Infant Vaccines): Groups MenACWY-CRM + Infant Vaccines (US1 +US3) pooled.
  US infants received MenACWY at 2, 4 and 6 months of age along with routine infant vaccines, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccine. These infants either received a fourth dose of MenACWY concomitantly with pneumococcal, HAV, and MMR-V vaccines at 12 months of age (US1A and US3) or received pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months and a fourth dose of MenACWY at 13 months of age( US1B).
- US2 + US4 (Infant Vaccines Only): Groups Infant Vaccines only (US2+US4) pooled
  US infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. These infants received:
  either one dose of MenACWY concomitantly with pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and a second dose of MenACWY at 15 months of age (US2 and US4A); or received concomitant pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months and one dose of MenACWY at 13 and one dose at 15 months of age (US4B); or one dose of MenACWY at 18 months of age (US4C).
- LA3 + LA5 (Men ACWY-CRM + Infant Vaccines): Groups Men ACWY-CRM + Infant Vaccines (LA3 and LA5) pooled.
  LA infants received MenACWY at 2, 4 and 6 months of age; and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines. At 12 months of age these infants were:
  1. Recommended to receive pneumococcal conjugate vaccine, HAV, and MMR-V. At 16 months of age, these subjects received the fourth dose of MenACWY along with concomitant DTaP and Hib (LA3A)
  2. Received pneumococcal conjugate vaccine, HAV, and MMR-V. At 16 months of age, these subjects received DTaP and Hib. At 17 months of age, these subjects received the fourth dose of MenACWY (LA3B).
  3. Received the fourth dose of MenACWY concomitantly with pneumococcal conjugate vaccine, HAV, and MMR-V (LA5).
- LA4 + LA6 (Infant Vaccines Only): Groups Infant Vaccines only (LA4 and LA6) pooled.
  LA infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus, and pneumococcal conjugate vaccines, at 2, 4 and 6 months of age. These infants received either:
  1. One dose of MenACWY concomitantly with pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months and a second dose of MenACWY along with DTaP and Hib vaccines at 15 months of age (LA4).
  2. Concomitant pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and either one dose each of MenACWY at 12 and 15 months of age (LA6A); or one dose each of MenACWY at 13 and 15 months of age (LA6B) or one dose of MenACWY at 18 months of age (LA6C).
Arm/Group | US1 + US3 (Men ACWY-CRM + Infant Vaccines) | US2 + US4 (Infant Vaccines Only) | LA3 + LA5 (Men ACWY-CRM + Infant Vaccines) | LA4 + LA6 (Infant Vaccines Only)
Number analyzed (Participants) | 989 | 503 | 1724 | 859
Subjects
  Erythema (mm) - Any | 93 | 77 | 628 | 338
  Erythema (mm) - Severe | 0 | 6 | 2 | 5
  Induration (mm) - Any | 85 | 69 | 321 | 179
  Induration (mm) - Severe | 0 | 1 | 2 | 0
  Tenderness - Any | 464 | 230 | 1086 | 596
  Tenderness - Severe | 32 | 25 | 114 | 94
  Body Temp. ( >= 38° C ) | 51 | 28 | 229 | 102
  Change in Eating Habits - Any | 259 | 130 | 294 | 143
  Change in Eating Habits - Severe | 10 | 3 | 6 | 5
  Diarrhea - Any | 154 | 63 | 266 | 118
  Diarrhea - Severe | 5 | 2 | 3 | 2
  Irritability - Any | 608 | 307 | 607 | 299
  Irritability - Severe | 32 | 16 | 26 | 4
  Persistent Crying - Any | 369 | 174 | 566 | 301
  Persistent Crying - Severe | 14 | 13 | 40 | 29
  Rash - Any | 31 | 16 | 110 | 59
  Rash - Severe | 11 | 6 | 58 | 27
  Sleepiness - Any | 541 | 249 | 820 | 433
  Sleepiness - Severe | 19 | 3 | 27 | 18
  Vomiting - Any | 100 | 50 | 244 | 117
  Vomiting - Severe | 0 | 1 | 3 | 2
  Analgesic / Antipyretic medication used | 672 | 333 | 1155 | 590

10. Secondary Outcome: Number of Subjects With Solicited Local and Systemic Reactions Post Second Vaccination - Infant Series
Description: Solicited local and systemic reactions reported post second vaccination was compared in subjects receiving MenACWY versus Hib Vaccines.
Time Frame: 7 days post-vaccination
Population: The population used in analysis was the safety set: The total number of subjects analyzed was less than the safety set due to subject withdrawals. Only subjects who received the second dose of the infant series vaccination were included in the analysis.
Measure: Number; unit: Subjects
Groups:
- US1+US3 (Men ACWY-CRM + Infant Vaccines): Groups MenACWY-CRM + Infant Vaccines (US1 +US3) pooled. US infants received MenACWY at 2, 4 and 6 months of age along with routine infant vaccines, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccine. These infants either received a fourth dose of MenACWY concomitantly with pneumococcal, HAV, and MMR-V vaccines at 12 months of age (US1A and US3) or received pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months and a fourth dose of MenACWY at 13 months of age( US1B).
- US2+US4 (Infant Vaccines Only): Groups Infant Vaccines only (US2+US4) pooled US infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. These infants received either one dose of MenACWY concomitantly with pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and a second dose of MenACWY at 15 months of age (US2 and US4A) or received concomitant pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months and one dose of MenACWY at 13 and a second dose of MenACWY at 15 months of age (US4B) or one dose of MenACWY at 18 months of age (US4C).
- LA3+LA5 (Men ACWY-CRM + Infant Vaccines): LA infants received MenACWY at 2, 4 and 6 months of age; and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines. At 12 months of age these infants were:
  1. Recommended to receive pneumococcal conjugate vaccine, HAV, and MMR-V. At 16 months of age, these subjects received the fourth dose of MenACWY along with concomitant DTaP and Hib (LA3A)
  2. Received pneumococcal conjugate vaccine, HAV, and MMR-V. At 16 months of age, these subjects received DTaP and Hib. At 17 months of age, these subjects received the fourth dose of MenACWY (LA3B).
  3. Received the fourth dose of MenACWY concomitantly with pneumococcal conjugate vaccine, HAV, and MMR-V (LA5).
- LA4+LA6 (Infant Vaccines Only): Groups Infant Vaccines only (LA4 and LA6) pooled.
  LA infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus, and pneumococcal conjugate vaccines, at 2, 4 and 6 months of age. These infants received either:
  1. One dose of MenACWY concomitantly with pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months and a second dose of MenACWY along with DTaP and Hib vaccines at 15 months of age (LA4).
  2. Concomitant pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and either one dose each of MenACWY at 12 and 15 months of age (LA6A); or one dose each of MenACWY at 13 and 15 months of age (LA6B) or one dose of MenACWY at 18 months of age (LA6C).
Arm/Group | US1+US3 (Men ACWY-CRM + Infant Vaccines) | US2+US4 (Infant Vaccines Only) | LA3+LA5 (Men ACWY-CRM + Infant Vaccines) | LA4+LA6 (Infant Vaccines Only)
Number analyzed (Participants) | 936 | 476 | 1672 | 824
Subjects
  Erythema (mm) - Any | 108 | 95 | 675 | 356
  Erythema (mm) - Severe | 0 | 2 | 0 | 0
  Induration (mm) - Any | 77 | 75 | 267 | 162
  Induration (mm) - Severe | 1 | 3 | 0 | 0
  Tenderness - Any | 348 | 193 | 841 | 460
  Tenderness - Severe | 14 | 13 | 62 | 50
  Body Temp. ( >= 38° C ) | 72 | 43 | 246 | 135
  Change in Eating Habits - Any | 168 | 84 | 188 | 102
  Change in Eating Habits - Severe | 3 | 0 | 9 | 5
  Diarrhea - Any | 79 | 46 | 177 | 104
  Diarrhea - Severe | 2 | 3 | 5 | 1
  Irritability - Any | 505 | 265 | 496 | 250
  Irritability - Severe | 16 | 12 | 16 | 5
  Persistent Crying - Any | 261 | 141 | 336 | 209
  Persistent Crying - Severe | 5 | 4 | 18 | 11
  Rash - Any | 32 | 17 | 110 | 48
  Rash - Severe | 10 | 5 | 57 | 30
  Sleepiness - Any | 363 | 178 | 547 | 263
  Sleepiness - Severe | 3 | 3 | 17 | 8
  Vomiting - Any | 66 | 34 | 156 | 85
  Vomiting - Severe | 0 | 1 | 4 | 0
  Analgesic / Antipyretic medication used | 570 | 297 | 988 | 491

11. Secondary Outcome: Number of Subjects With Solicited Local and Systemic Reactions Post Third Vaccination - Infant Series
Description: Solicited local and systemic reactions reported post third vaccination was compared in subjects receiving MenACWY versus Hib Vaccines.
Time Frame: 7 days post-vaccination
Population: The population used in analysis was the safety set: The total number of subjects analyzed was less than the safety set due to subject withdrawals. Only subjects who received the third dose in the infant series were included in this analysis.
Measure: Number; unit: Subjects
Groups:
- US2+US4 (Infant Vaccines Only): Groups Infant Vaccines only (US2+US4) pooled US infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. These infants received either one dose of MenACWY concomitantly with pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and a second dose of MenACWY at 15 months of age (US2 and US4A) or received concomitant pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months and one dose of MenACWY at 13 and and a second dose of MenACWY at 15 months of age (US4B) or one dose of MenACWY at 18 months of age (US4C).
- LA3+LA5 (Men ACWY-CRM + Infant Vaccines): Groups Men ACWY-CRM + Infant Vaccines (LA3 and LA5) pooled
  LA infants received MenACWY at 2, 4 and 6 months of age; and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines. At 12 months of age these infants were:
  1. Recommended to receive pneumococcal conjugate vaccine, HAV, and MMR-V. At 16 months of age, these subjects received the fourth dose of MenACWY along with concomitant DTaP and Hib (LA3A)
  2. Received pneumococcal conjugate vaccine, HAV, and MMR-V. At 16 months of age, these subjects received DTaP and Hib. At 17 months of age, these subjects received the fourth dose of MenACWY (LA3B).
  3. Received the fourth dose of MenACWY concomitantly with pneumococcal conjugate vaccine, HAV, and MMR-V (LA5).
Arm/Group | US1+US3 (Men ACWY-CRM + Infant Vaccines) | US2+US4 (Infant Vaccines Only) | LA3+LA5 (Men ACWY-CRM + Infant Vaccines) | LA4+LA6 (Infant Vaccines Only)
Number analyzed (Participants) | 910 | 454 | 1646 | 826
Subjects
  Erythema (mm) - Any | 126 | 95 | 549 | 311
  Erythema (mm) - Severe | 0 | 2 | 2 | 1
  Induration (mm) - Any | 89 | 82 | 189 | 105
  Induration (mm) - Severe | 0 | 3 | 1 | 0
  Tenderness - Any | 271 | 137 | 582 | 356
  Tenderness - Severe | 1 | 8 | 23 | 15
  Body Temp. ( >= 38° C ) | 46 | 34 | 190 | 115
  Change in Eating Habits - Any | 135 | 57 | 149 | 75
  Change in Eating Habits - Severe | 3 | 3 | 6 | 3
  Diarrhea - Any | 63 | 35 | 109 | 69
  Diarrhea - Severe | 2 | 1 | 2 | 3
  Irritability - Any | 416 | 227 | 373 | 192
  Irritability - Severe | 6 | 6 | 7 | 2
  Persistent Crying - Any | 189 | 98 | 208 | 130
  Persistent Crying - Severe | 4 | 4 | 11 | 2
  Rash - Any | 25 | 12 | 68 | 30
  Rash - Severe | 7 | 4 | 32 | 11
  Sleepiness - Any | 257 | 130 | 362 | 181
  Sleepiness - Severe | 6 | 1 | 7 | 3
  Vomiting - Any | 43 | 29 | 115 | 64
  Vomiting - Severe | 0 | 1 | 2 | 1
  Analgesic / Antipyretic medication used | 506 | 274 | 682 | 393

12. Secondary Outcome: Geometric Mean hSBA Titers Post-infant Series - US Subjects
Description: Geometric Mean hSBA Titers directed against N. meningitidis serogroups A, C, W and Y was measured after three doses at 2, 4, and 6 months of age.
Time Frame: 7 months of age (one month post-infant series)
Population: The analysis was done on per protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- US1 (MenACWY-CRM + Infant Vaccines): US infants received one dose of MenACWY at 2, 4 and 6 months of age and received,as part of routine infant vaccination schedule, DTaP-IPV-HBV, Hib, pneumococcal conjugate vaccine, and rotavirus vaccine. Group US1 was randomized into subgroups US1A and US1B.
- US2 (Infant Vaccines Only): received as part of routine infant vaccination schedule DTaP-IPV-HBV,Hib, pneumococcal conjugate vaccine, and rotavirus vaccine at 2, 4 and 6 months of age. At 12 months of age, these subjects received a dose of MenACWY along with concomitant pneumococcal conjugate vaccine, HAV, and MMR-V. At 15 months of age, these subjects received a second dose of MenACWY.
Arm/Group | US1 (MenACWY-CRM + Infant Vaccines) | US2 (Infant Vaccines Only)
Number analyzed (Participants) | 212 | 90
Titers
  A (Pre-vaccination GMT; N= 177, 65) | 2.11 [2 to 2.23] | 2.1 [1.92 to 2.29]
  A (Post-vaccination GMT; N= 212, 80) | 13 [11 to 16] | 2.03 [1.53 to 2.7]
  C (Pre-vaccination GMT; N= 168, 64) | 2.48 [2.23 to 2.75] | 2.17 [1.83 to 2.57]
  C (Post-vaccination GMT; N= 204, 84) | 108 [92 to 127] | 2.12 [1.64 to 2.74]
  W (Pre-vaccination GMT; N= 165, 66) | 3.07 [2.7 to 3.5] | 2.71 [2.2 to 3.33]
  W (Post-vaccination GMT; N=197, 90) | 100 [86 to 116] | 2.08 [1.67 to 2.6]
  Y (Pre-vaccination GMT; N=150, 62 ) | 2.53 [2.31 to 2.77] | 2.13 [1.85 to 2.45]
  Y (Post-vaccination GMT; N=182, 84) | 73 [62 to 86] | 2.03 [1.6 to 2.57]

13. Secondary Outcome: Geometric Mean hSBA Titers Post-infant Series - LA Subjects
Description: Geometric Mean hSBA Titers directed against N. meningitidis serogroups A, C, W and Y was measured after two doses of MenACWY at 2 and 6 months (LA1) versus three doses at 2, 4, and 6 (LA3) months of age.
Time Frame: 7 months of age (one month post-infant series)
Population: Per protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | LA1 (MenACWY-CRM + Infant Vaccines) | LA3 (MenACWY-CRM + Infant Vaccines)
Number analyzed (Participants) | 277 | 272
Titer
  A (Pre-vaccination GMT; N= 272, 271) | 2.09 [2.03 to 2.16] | 2.03 [1.97 to 2.09]
  A (Post-vaccination GMT; N= 277, 268) | 31 [26 to 38] | 43 [36 to 52]
  C (Pre-vaccination GMT; N= 273,272) | 2.32 [2.18 to 2.47] | 2.34 [2.19 to 2.49]
  C (Post-vaccination GMT; N= 277, 272) | 155 [131 to 183] | 150 [127 to 177]
  W (Pre-vaccination GMT; N= 263, 261) | 2.9 [2.64 to 3.18] | 2.54 [2.31 to 2.79]
  W (Post-vaccination GMT; N=271,264) | 259 [227 to 296] | 182 [159 to 208]
  Y (Pre-vaccination GMT; N=258, 260) | 2.35 [2.22 to 2.49] | 2.26 [2.14 to 2.39]
  Y (Post-vaccination GMT; N=272,263) | 159 [136 to 185] | 125 [107 to 146]
Statistical Analysis 1: Comparison: LA1 (MenACWY-CRM + Infant Vaccines) vs LA3 (MenACWY-CRM + Infant Vaccines); Serogroup A (Post-vaccination GMT; group ratio LA1:LA3); Test type: Non-Inferiority or Equivalence — LA1 was noninferior to LA3, if the lower limit of the two-sided 95% CI for the ratio of GMTs between the 2 dose and the 3 dose schedule (GMTLA1/GMTLA3) must be > 0.5; ANOVA; Ratio of GMT = 0.73, 95% CI 2-sided [0.55 to 0.95]
Statistical Analysis 2: Comparison: LA1 (MenACWY-CRM + Infant Vaccines) vs LA3 (MenACWY-CRM + Infant Vaccines); Serogroup C (Post-vaccination GMT; group ratio LA1:LA3); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; ANOVA; Ratio of GMTs = 1.03, 95% CI 2-sided [0.81 to 1.31]
Statistical Analysis 3: Comparison: LA1 (MenACWY-CRM + Infant Vaccines) vs LA3 (MenACWY-CRM + Infant Vaccines); Serogroup W (Post-vaccination GMT; group ratio LA1:LA3); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; ANOVA; Ratio of GMTs = 1.42, 95% CI 2-sided [1.18 to 1.72]
Statistical Analysis 4: Comparison: LA1 (MenACWY-CRM + Infant Vaccines) vs LA3 (MenACWY-CRM + Infant Vaccines); Serogroup Y (Post-vaccination GMT; group ratio LA1:LA3); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 13, analysis 1]; ANOVA; Ratio of GMTs = 1.27, 95% CI 2-sided [1.02 to 1.58]

14. Secondary Outcome: Percentage of Subjects With hSBA Titer >=1:8 - US Subjects
Description: Immunogenicity as measured by percentage of subjects with hSBA titer >=1:8 directed against N. meningitidis serogroups A, C, W and Y; after three doses of MenACWY at 2, 4, and 6 months of age.
Time Frame: 7 months of age (one month post-infant series)
Population: Per Protocol Population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | US1 (MenACWY-CRM + Infant Vaccines) | US2 (Infant Vaccines Only)
Number analyzed (Participants) | 212 | 90
Percentages of subjects
  A (Pre-vaccination GMT; N= 177, 65) | 2 [0 to 5] | 3 [0 to 11]
  A (Post-vaccination GMT; N= 212, 80) | 67 [61 to 74] | 1 [0.032 to 7]
  C (Pre-vaccination GMT; N= 168, 64) | 7 [3 to 11] | 5 [1 to 13]
  C (Post-vaccination GMT; N= 204, 84) | 97 [93 to 99] | 1 [0.03 to 6]
  W (Pre-vaccination GMT; N= 165, 66) | 17 [12 to 24] | 11 [4 to 21]
  W (Post-vaccination GMT; N=197, 90) | 96 [93 to 99] | 2 [0 to 8]
  Y (Pre-vaccination GMT; N=150, 62 ) | 5 [2 to 10] | 3 [0 to 11]
  Y (Post-vaccination GMT; N=182, 84) | 96 [92 to 98] | 0 [0 to 4]

15. Secondary Outcome: Percentage of Subjects With hSBA Titer >=1:4 - US Subjects
Description: Immunogenicity as measured by percentage of subjects with hSBA titer >=1:4 directed against N. meningitidis serogroups A, C, W and Y; after three doses of MenACWY at 2, 4, and 6 months of age.
Time Frame: 7 months of age (one month post-infant series)
Population: Per Protocol Population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | US1 (MenACWY-CRM + Infant Vaccines) | US2 (Infant Vaccines Only)
Number analyzed (Participants) | 212 | 90
Percentages of subjects
  A (Pre-vaccination GMT; N= 177, 65) | 2 [1 to 6] | 3 [0 to 11]
  A (Post-vaccination GMT; N= 212, 80) | 71 [65 to 77] | 1 [0.03 to 7]
  C (Pre-vaccination GMT; N= 168, 64) | 10 [6 to 16] | 5 [1 to 13]
  C (Post-vaccination GMT; N= 204, 84) | 99 [96 to 100] | 2 [0 to 8]
  W (Pre-vaccination GMT; N= 165, 66) | 22 [16 to 30] | 15 [8 to 26]
  W (Post-vaccination GMT; N=197, 90) | 99 [96 to 100] | 2 [0 to 8]
  Y (Pre-vaccination GMT; N=150, 62 ) | 17 [11 to 24] | 5 [1 to 13]
  Y (Post-vaccination GMT; N=182, 84) | 98 [98 to 100] | 1 [0.032 to 6]

16. Secondary Outcome: Percentage of Subjects With hSBA Titer >=1:8 - LA Subjects
Description: Immunogenicity as measured by percentage of subjects with hSBA titer >=1:8 directed against N. meningitidis serogroups A, C, W and Y; after two doses of MenACWY at 2 and 6 months (LA1) versus three doses at 2, 4, and 6 months of age (LA3) .
Time Frame: 7 months of age (one month post-infant series)
Population: Per protocol population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | LA1 (MenACWY-CRM + Infant Vaccines) | LA3 (MenACWY-CRM + Infant Vaccines)
Number analyzed (Participants) | 277 | 272
Percentages of subjects
  A (Pre-vaccination hSBA titer ≥1:8; N= 272, 271) | 1 [0 to 4] | 0 [0 to 2]
  A (Post-vaccination hSBA titer ≥1:8; N= 277, 268) | 74 [69 to 79] | 89 [85 to 93]
  C (Pre-vaccination hSBA titer ≥1:8; N= 273,272) | 4 [2 to 7] | 4 [2 to 8]
  C (Post-vaccination hSBA titer ≥1:8; N= 277, 272) | 94 [90 to 96] | 97 [94 to 99]
  W (Pre-vaccination hSBA titer ≥1:8; N= 263, 261) | 16 [12 to 21] | 10 [7 to 14]
  W (Post-vaccination hSBA titer ≥1:8; N=271,264) | 99 [97 to 100] | 98 [96 to 100]
  Y (Pre-vaccination hSBA titer ≥1:8; N=258, 260) | 5 [3 to 9] | 3 [2 to 6]
  Y (Post-vaccination hSBA titer ≥1:8; N=272,263) | 97 [94 to 99] | 98 [96 to 99]
Statistical Analysis 1: Comparison: LA1 (MenACWY-CRM + Infant Vaccines) vs LA3 (MenACWY-CRM + Infant Vaccines); Serogroup A (post-vaccination percentage of subjects with hSBA titer >=8, group difference (PLA1 - PLA3)); Test type: Non-Inferiority or Equivalence — LA1 was noninferior to LA3, if the lower limit of the two-sided 95% CI for the difference in percentage of subjects with hSBA ≥ 1:8 and ≥1:4 between the 2 dose and the 3 dose schedule (PLA1 - PLA3) must be greater than -10%; ANOVA; Percentage (hSBA titers >=8) difference = -15, 95% CI 2-sided [-21.2 to -8.5]
Statistical Analysis 2: Comparison: LA1 (MenACWY-CRM + Infant Vaccines) vs LA3 (MenACWY-CRM + Infant Vaccines); Serogroup C (post-vaccination percentage of subjects with hSBA titer >=8, group difference (PLA1 - PLA3)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 16, analysis 1]; ANOVA; Percentage (hSBA titers >=8) difference = -3, 95% CI 2-sided [-7 to 0.3]
Statistical Analysis 3: Comparison: LA1 (MenACWY-CRM + Infant Vaccines) vs LA3 (MenACWY-CRM + Infant Vaccines); Serogroup W (post-vaccination percentage of subjects with hSBA titer >=8, group difference (PLA1 - PLA3)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 16, analysis 1]; ANOVA; Percentage (hSBA titers >=8) difference = 1, 95% CI 2-sided [-1.3 to 3.1]
Statistical Analysis 4: Comparison: LA1 (MenACWY-CRM + Infant Vaccines) vs LA3 (MenACWY-CRM + Infant Vaccines); Serogroup Y (post-vaccination percentage of subjects with hSBA titer >=8, group difference (PLA1 - PLA3)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 16, analysis 1]; ANOVA; Percentage (hSBA titers >=8) difference = -1, 95% CI 2-sided [-4 to 1.7]

17. Secondary Outcome: Percentage of Subjects With hSBA Titer >=1:4 - LA Subjects
Description: Immunogenicity as measured by percentage of subjects with hSBA titer >=1:4 directed against N. meningitidis serogroups A, C, W and Y; after two doses of MenACWY at 2 and 6 months (LA1) versus three doses at 2, 4, and 6 months of age (LA3) .
Time Frame: 7 months of age (one month post-infant series)
Population: Per protocol population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | LA1 (MenACWY-CRM + Infant Vaccines) | LA3 (MenACWY-CRM + Infant Vaccines)
Number analyzed (Participants) | 277 | 272
Percentages of subjects
  A (Pre-vaccination hSBA titer ≥1:4; N= 272, 271) | 2 [1 to 5] | 1 [0 to 3]
  A (Post-vaccination hSBA titer ≥1:4; N= 277, 268) | 78 [73 to 83] | 91 [87 to 94]
  C (Pre-vaccination hSBA titer ≥1:4; N= 273,272) | 10 [7 to 14] | 10 [7 to 15]
  C (Post-vaccination hSBA titer ≥1:4; N= 277, 272) | 96 [93 to 98] | 98 [96 to 99]
  W (Pre-vaccination hSBA titer ≥1:4; N= 263, 261) | 17 [13 to 23] | 13 [9 to 17]
  W (Post-vaccination hSBA titer ≥1:4; N=271,264) | 100 [99 to 100] | 99 [97 to 100]
  Y (Pre-vaccination hSBA titer ≥1:4; N=258, 260) | 11 [8 to 16] | 8 [5 to 13]
  Y (Post-vaccination hSBA titer ≥1:4; N=272,263) | 98 [96 to 99] | 99 [97 to 100]

18. Secondary Outcome: Geometric Mean Concentrations or Titers of DTaP, HBV, Hib, Pneumococcal and Polio Antigens at 1 Month After Infant Series Vaccination - US Subjects
Description: Immunogenicity as measured by antibody GMCs / GMTs directed against DTaP, HBV, Hib, pneumococcal and polio antigens.
Time Frame: 7 months of age (one month post-infant series)
Population: Per Protocol
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- US1 (Men ACWY-CRM + Infant Vaccines): US infants received one dose of MenACWY at 2, 4 and 6 months of age; and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines. Group US1 was randomized into US1A and US1B subgroups.
Arm/Group | US1 (Men ACWY-CRM + Infant Vaccines) | US2 (Infant Vaccines Only)
Number analyzed (Participants) | 214 | 102
Titers
  Diphtheria (214, 102) | 2.52 [2.28 to 2.78] | 2.88 [2.5 to 3.32]
  Tetanus (214, 102) | 2.5 [2.28 to 2.74] | 2.31 [2.01 to 2.64]
  PT (174, 83) | 54 [48 to 62] | 54 [44 to 66]
  FHA (174, 83) | 118 [106 to 132] | 114 [97 to 134]
  Pertactin (174, 83) | 114 [100 to 130] | 110 [90 to 134]
  Polio Type 1 (176, 98) | 422 [363 to 491] | 441 [361 to 540]
  Polio Type 2 (175, 98) | 348 [297 to 408] | 290 [235 to 358]
  Polio Type 3 (176, 98) | 733 [607 to 885] | 635 [493 to 818]
  Hepatitis B (N=148, N=98) | 1863 [1538 to 2257] | 2112 [1668 to 2674]
  Hib (N=213, N=101) | 4.64 [3.9 to 5.53] | 3.56 [2.77 to 4.58]
  PnC 4 (N=181, N=102) | 1.67 [1.5 to 1.86] | 2 [1.73 to 2.3]
  PnC 6B (N=181, N=102) | 1.94 [1.61 to 2.34] | 2.55 [1.99 to 3.27]
  PnC 9V (N=181, N=102) | 1.83 [1.62 to 2.06] | 2.15 [1.83 to 2.53]
  PnC 14 (N=181, N=102) | 6.97 [6.18 to 7.86] | 6.79 [5.78 to 7.96]
  PnC 18C (N=181, N=102) | 1.96 [1.75 to 2.19] | 2.54 [2.18 to 2.95]
  PnC 19F (N=181, N=102) | 2.24 [2.02 to 2.48] | 2.73 [2.39 to 3.13]
  PnC 23F (N=181, N=102) | 1.71 [1.47 to 1.98] | 2.15 [1.76 to 2.62]
Statistical Analysis 1: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); Diphtheria (Post-vaccination GMT; group ratio US1:US2); Test type: Non-Inferiority or Equivalence — To assess non-inferiority of US1 over US2, the lower limit of 95% CI for the ratio of pertussis GMCs (GMCUS1 /GMCUS2) must be greater than 0.67; the lower limit of 95% CI for the ratio of all other GMCs (GMCUS1 / GMCUS2) must be greater than 0.50; ANOVA; Ratio of GMTs = 0.87, 95% CI 2-sided [0.74 to 1.04]
Statistical Analysis 2: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); Tetanus (Post-vaccination GMT; group ratio US1:US2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 18, analysis 1]; ANOVA; Ratio of GMTs = 1.08, 95% CI 2-sided [0.92 to 1.28]
Statistical Analysis 3: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); PT (Post-vaccination GMT; group ratio US1:US2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 18, analysis 1]; ANOVA; Ratio of GMTs = 1, 95% CI 2-sided [0.79 to 1.26]
Statistical Analysis 4: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); FHA (Post-vaccination GMT; group ratio US1:US2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 18, analysis 1]; Ratio of GMTs = 1.03, 95% CI 2-sided [0.85 to 1.25]
Statistical Analysis 5: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); Pertactin (Post-vaccination GMT; group ratio US1:US2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 18, analysis 1]; ANOVA; Ratio of GMTs = 1.04, 95% CI 2-sided [0.83 to 1.32]
Statistical Analysis 6: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); Polio Type 1 (Post-vaccination GMT; group ratio US1:US2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 18, analysis 1]; ANOVA; Ratio of GMTs = 0.96, 95% CI 2-sided [0.75 to 1.23]
Statistical Analysis 7: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); Polio Type 2 (Post-vaccination GMT; group ratio US1:US2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 18, analysis 1]; ANOVA; Ratio of GMTs = 1.2, 95% CI 2-sided [0.93 to 1.55]
Statistical Analysis 8: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); Polio Type 3 (Post-vaccination GMT; group ratio US1:US2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 18, analysis 1]; ANOVA; Ratio of GMTs = 1.15, 95% CI 2-sided [0.85 to 1.56]
Statistical Analysis 9: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); Hepatitis B (Post-vaccination GMT; group ratio US1:US2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 18, analysis 1]; ANOVA; Ratio of GMTs = 0.88, 95% CI [0.65 to 1.2]
Statistical Analysis 10: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); HIb (Post-vaccination GMT; group ratio US1:US2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 18, analysis 1]; ANOVA; Ratio of GMTs = 1.31, 95% CI 2-sided [0.97 to 1.77]
Statistical Analysis 11: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); PnC 4 (Post-vaccination GMT; group ratio US1:US2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 18, analysis 1]; ANOVA; Ratio of GMTs = 0.84, 95% CI 2-sided [0.7 to 1]
Statistical Analysis 12: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); PnC 6B (Post-vaccination GMT; group ratio US1:US2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 18, analysis 1]; ANOVA; Ratio of GMTs = 0.76, 95% CI 2-sided [0.56 to 1.03]
Statistical Analysis 13: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); PnC 9V (Post-vaccination GMT; group ratio US1:US2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 18, analysis 1]; ANOVA; Ratio of GMTs = 0.85, 95% CI [0.7 to 1.04]
Statistical Analysis 14: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); PnC 14 (Post-vaccination GMT; group ratio US1:US2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 18, analysis 1]; ANOVA; Ratio of GMTs = 1.03, 95% CI 2-sided [0.84 to 1.26]
Statistical Analysis 15: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); PnC 18C (Post-vaccination GMT; group ratio US1:US2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 18, analysis 1]; ANOVA; Ratio of GMTs = 0.77, 95% CI 2-sided [0.64 to 0.93]
Statistical Analysis 16: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); PnC 19F (Post-vaccination GMT; group ratio US1:US2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 18, analysis 1]; ANOVA; Ratio of GMTs = 0.82, 95% CI 2-sided [0.69 to 0.97]
Statistical Analysis 17: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); PnC 23F (Post-vaccination GMT; group ratio US1:US2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 18, analysis 1]; ANOVA; Ratio of GMTs = 0.79, 95% CI 2-sided [0.62 to 1.02]

19. Secondary Outcome: Seroresponse Rates to DTaP, HBV, Hib, Pneumococcal and Polio Antigens at 1 Month After Infant Series Vaccination - US Subjects
Description: Immunogenicity as measured by percentage of subjects with predefined seroprotective antibody titers against DTaP, HBV, Hib, pneumococcal and polio antigens.
Time Frame: 7 months of age (one month post-infant series)
Population: Per Protocol
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | US1 (Men ACWY-CRM + Infant Vaccines) | US2 (Infant Vaccines Only)
Number analyzed (Participants) | 214 | 102
Percentages of subjects
  Diphtheria (≥ 0.1 IU/mL) (214, 102) | 100 [97 to 100] | 100 [96 to 100]
  Tetanus (≥ 0.1 IU/mL) (214, 102) | 100 [98 to 100] | 100 [96 to 100]
  PT(≥ 4-fold rise) (174, 83) | 87 [81 to 92] | 86 [76 to 92]
  FHA (≥ 4-fold rise) (174, 83) | 85 [79 to 90] | 80 [69 to 88]
  Pertactin (≥ 4-fold rise) (174, 83) | 76 [69 to 83] | 78 [68 to 87]
  Polio Type 1 (≥1:8) (176, 98) | 99 [97 to 100] | 100 [96 to 100]
  Polio Type 2 (≥1:8) (176, 98) | 100 [98 to 100] | 100 [96 to 100]
  Polio Type 3 (≥1:8)(175, 98) | 99 [97 to 100] | 100 [96 to 100]
  Hepatitis B (≥10 mIU/mL) (N=148, N=98) | 99 [96 to 100] | 100 [96 to 100]
  Hib (≥ 0.15 μg/mL) (N=213, N=101) | 99 [97 to 100] | 100 [96 to 100]
  Hib (≥1.0 μg/mL) (N=213, N=101) | 89 [84 to 93] | 84 [76 to 91]
  PnC 4 (≥ 0.35 μg/mL) (N=181, N=102) | 98 [95 to 100] | 100 [96 to 100]
  PnC 6B (≥ 0.35 μg/mL) (N=181, N=102) | 88 [83 to 93] | 96 [90 to 99]
  PnC 9V (≥ 0.35 μg/mL) (N=181, N=102) | 98 [94 to 99] | 98 [93 to 100]
  PnC 14 (≥ 0.35 μg/mL) (N=181, N=102) | 100 [98 to 100] | 99 [95 to 100]
  PnC 18C (≥ 0.35 μg/mL) (N=181, N=102) | 97 [94 to 99] | 100 [96 to 100]
  PnC 19F (≥ 0.35 μg/mL) (N=181, N=102) | 99 [96 to 100] | 100 [96 to 100]
  PnC 23F (≥ 0.35 μg/mL) (N=181, N=102) | 92 [87 to 95] | 94 [88 to 98]
Statistical Analysis 1: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); Diphtheria (Seroconversion percentage difference (PUS1 - PUS2)); Test type: Non-Inferiority or Equivalence — To assess non-inferiority of US1 over US2, the lower limit of 95% CI for the difference in seroresponse rates (PUS1 - PUS2) must be greater than -5% for polio and -10% for all others; ANOVA; Seroconversion Percentage difference = 0, 95% CI 2-sided [-3 to 3]
Statistical Analysis 2: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); Tetanus (Seroconversion percentage difference (PUS1 - PUS2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 1]; ANOVA; Seroconversion Percentage difference = 0, 95% CI 2-sided [-2 to 4]
Statistical Analysis 3: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); PT (Seroconversion percentage difference (PUS1 - PUS2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 1]; ANOVA; Seroconversion Percentage difference = 2, 95% CI 2-sided [-7 to 12]
Statistical Analysis 4: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); FHA(Seroconversion percentage difference (PUS1 - PUS2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 1]; ANOVA; Seroconversion Percentage difference = 6, 95% CI 2-sided [-4 to 17]
Statistical Analysis 5: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); Pertactin (Seroconversion percentage difference (PUS1 - PUS2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 1]; ANOVA; Seroconversion Percentage difference = -2, 95% CI 2-sided [-12 to 10]
Statistical Analysis 6: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); Polio Type 1 (Seroconversion percentage difference (PUS1 - PUS2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 1]; ANOVA; Seroconversion Percentage difference = -1, 95% CI 2-sided [-3 to 3]
Statistical Analysis 7: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); Polio Type 2 (Seroconversion percentage difference (PUS1 - PUS2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 1]; ANOVA; Seroconversion Percentage difference = 0, 95% CI 2-sided [-2 to 4]
Statistical Analysis 8: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); Polio Type 3 (Seroconversion percentage difference (PUS1 - PUS2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 1]; ANOVA; Seroconversion Percentage difference = -1, 95% CI 2-sided [-3 to 3]
Statistical Analysis 9: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); Hepatitis B(Seroconversion percentage difference (PUS1 - PUS2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 1]; ANOVA; Seroconversion Percentage difference = -1, 95% CI 2-sided [-4 to 3]
Statistical Analysis 10: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); Hib (≥ 0.15 μg/mL)(Seroconversion percentage difference (PUS1 - PUS2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 1]; ANOVA; Seroconversion Percentage difference = -1, 95% CI 2-sided [-3 to 3]
Statistical Analysis 11: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); Hib (≥1.0 μg/mL)(Seroconversion percentage difference (PUS1 - PUS2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 1]; ANOVA; Seroconversion Percentage difference = 5, 95% CI 2-sided [-3 to 14]
Statistical Analysis 12: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); PnC 4(Seroconversion percentage difference (PUS1 - PUS2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 1]; ANOVA; Seroconversion Percentage difference = -2, 95% CI 2-sided [-5 to 2]
Statistical Analysis 13: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); PnC 6B(Seroconversion percentage difference (PUS1 - PUS2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 1]; ANOVA; (Seroconversion percentage difference (P = -8, 95% CI 2-sided [-14 to -1]
Statistical Analysis 14: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); PnC 9V (Seroconversion percentage difference (PUS1 - PUS2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 1]; ANOVA; Seroconversion Percentage difference = 0, 95% CI 2-sided [-4 to 5]
Statistical Analysis 15: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); PnC 14 (Seroconversion percentage difference (PUS1 - PUS2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 1]; ANOVA; Diphtheria (Seroconversion percentage di = 1, 95% CI 2-sided [-1 to 5]
Statistical Analysis 16: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); PnC 18C (Seroconversion percentage difference (PUS1 - PUS2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 1]; ANOVA; Seroconversion Percentage difference = -3, 95% CI 2-sided [-6 to 1]
Statistical Analysis 17: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); PnC 19F (Seroconversion percentage difference (PUS1 - PUS2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 1]; ANOVA; (Seroconversion percentage difference (P = -1, 95% CI 2-sided [-4 to 3]
Statistical Analysis 18: Comparison: US1 (Men ACWY-CRM + Infant Vaccines) vs US2 (Infant Vaccines Only); PnC 23F (Seroconversion percentage difference (PUS1 - PUS2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 1]; ANOVA; Seroconversion Percentage difference = -2, 95% CI 2-sided [-8 to 5]

20. Secondary Outcome: Geometric Mean Concentrations or Titers of DTaP, HBV, Hib, Pneumococcal and Polio Antigens at 1 Month After Infant Series Vaccination - LA Subjects
Description: Immunogenicity as measured by antibody GMCs / GMTs directed against DTaP, HBV, Hib, pneumococcal and polio antigens.
Time Frame: 7 months of age (one month post-infant series)
Population: Per Protocol
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- LA1 (Men ACWY-CRM + Infant Vaccines): LA infants received MenACWY at 2 and 6 months of age and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. Group LA1 was randomized into LA1A and LA 1B subgroups.
- LA3 (Men ACWY-CRM + Infant Vaccines): LA infants received MenACWY at 2, 4 and 6 months of age; and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, pneumococcal conjugate vaccine, and rotavirus vaccine. Group LA3 was further randomized into LA3A and LA3B subgroups.
Arm/Group | LA1 (Men ACWY-CRM + Infant Vaccines) | LA2 (Infant Vaccines Only) | LA3 (Men ACWY-CRM + Infant Vaccines) | LA4 (Infant Vaccines Only)
Number analyzed (Participants) | 287 | 123 | 283 | 137
Titers
  Diphtheria (N=287, N=123, N=283, N=137) | 1.8 [1.62 to 1.99] | 1.54 [1.32 to 1.81] | 1.45 [1.31 to 1.61] | 1.77 [1.52 to 2.05]
  Tetanus (N=287, N=123, N=283, N=137) | 2.41 [2.23 to 2.6] | 2.19 [1.94 to 2.46] | 2.51 [2.33 to 2.71] | 2.65 [2.37 to 2.96]
  PT (N=285, N=123, N=281, N=135) | 47 [43 to 52] | 45 [39 to 53] | 45 [41 to 50] | 49 [42 to 56]
  FHA (N=286, N=123, N=281, N=135) | 102 [93 to 112] | 97 [85 to 112] | 99 [91 to 109] | 112 [99 to 128]
  Pertactin (N=286, N=123, N=281, N=135) | 123 [110 to 137] | 124 [105 to 146] | 119 [106 to 133] | 149 [127 to 175]
  Polio Type 1 (N=265, N=112, N=252, N=120) | 535 [462 to 620] | 598 [477 to 749] | 533 [458 to 619] | 684 [550 to 850]
  Polio Type 2 (N=265, N=112, N=252, N=120) | 353 [302 to 411] | 366 [289 to 463] | 318 [271 to 372] | 385 [306 to 483]
  Polio Type 3 (N=265, N=112, N=252, N=120) | 710 [596 to 846] | 747 [571 to 977] | 656 [548 to 785] | 813 [627 to 1054]
  Hepatitis B (N=243, N=104, N=237, N=118) | 2273 [2001 to 2583] | 2045 [1682 to 2485] | 1900 [1670 to 2162] | 1993 [1660 to 2394]
  Hib (N=287, N=123, N=283, N=137) | 7.64 [6.63 to 8.8] | 6.01 [4.84 to 7.47] | 7.19 [6.23 to 8.29] | 6.74 [5.49 to 8.28]
  PnC 4 (N=268, N=116, N=256, N=126) | 2.07 [1.88 to 2.27] | 2.24 [1.94 to 2.58] | 1.91 [1.74 to 2.1] | 2.39 [2.08 to 2.74]
  PnC 6B (N=264, N=116, N=255, N=124) | 2.15 [1.85 to 2.49] | 2.21 [1.76 to 2.77] | 2.09 [1.8 to 2.44] | 2.4 [1.93 to 2.98]
  PnC 9V (N=268, N=116, N=256, N=126) | 1.89 [1.71 to 2.1] | 2.21 [1.89 to 2.6] | 1.81 [1.63 to 2.02] | 2.19 [1.88 to 2.55]
  PnC 14 (N=268, N=116, N=256, N=126) | 7.29 [6.42 to 8.29] | 8.06 [6.63 to 9.78] | 7.69 [6.75 to 8.77] | 9.18 [7.62 to 11]
  PnC 18C (N=268, N=116, N=256, N=126) | 1.86 [1.68 to 2.07] | 2.09 [1.78 to 2.44] | 1.7 [1.53 to 1.89] | 2.26 [1.94 to 2.62]
  PnC 19F (N=268, N=116, N=254, N=126) | 2.34 [2.1 to 2.6] | 2.6 [2.2 to 3.06] | 2.3 [2.06 to 2.57] | 2.53 [2.16 to 2.96]
  PnC 23F (N=267, N=115, N=256, N=125) | 1.88 [1.64 to 2.16] | 2.46 [1.99 to 3.03] | 2.12 [1.84 to 2.44] | 2.42 [1.98 to 2.96]
Statistical Analysis 1: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); Diphtheria (Post-vaccination GMC; group ratio LA1:LA2); Test type: Non-Inferiority or Equivalence — To assess non-inferiority of LA1 to LA2, the lower limit of the 95% CI for the ratio of pertussis GMCs (GMCLA1 / GMCLA2) must be greater than 0.67; the lower limit of the 95% CI for the ratio of all other GMCs (GMCLA1 / GMCLA2) must be greater than 0.50; ANOVA; Ratio of GMCs = 1.16, 95% CI 2-sided [0.96 to 1.4]
Statistical Analysis 2: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); Tetanus (Post-vaccination GMC; group ratio LA1:LA2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 1]; ANOVA; Ratio of GMCs = 1.1, 95% CI 2-sided [0.96 to 1.27]
Statistical Analysis 3: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); PT (Post-vaccination GMC; group ratio LA1:LA2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 1]; ANOVA; Ratio of GMCs = 1.04, 95% CI 2-sided [0.87 to 1.25]
Statistical Analysis 4: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); FHA (Post-vaccination GMC; group ratio LA1:LA2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 1]; ANOVA; Ratio of GMCs = 1.05, 95% CI 2-sided [0.89 to 1.23]
Statistical Analysis 5: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); Pertactin (Post-vaccination GMC; group ratio LA1:LA2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 1]; ANOVA; Ratio of GMCs = 0.99, 95% CI 2-sided [0.81 to 1.21]
Statistical Analysis 6: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); Polio Type 1 (Post-vaccination GMT; group ratio LA1:LA2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 1]; ANOVA; Ratio of GMTs = 0.9, 95% CI 2-sided [0.68 to 1.17]
Statistical Analysis 7: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); Polio Type 2 (Post-vaccination GMT; group ratio LA1:LA2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 1]; ANOVA; Ratio of GMTs = 0.97, 95% CI 2-sided [0.73 to 1.28]
Statistical Analysis 8: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); Polio Type 3 (Post-vaccination GMT; group ratio LA1:LA2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 1]; ANOVA; Ratio of GMTs = 0.95, 95% CI [0.69 to 1.31]
Statistical Analysis 9: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); Hepatitis B (Post-vaccination GMC; group ratio LA1:LA2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 1]; ANOVA; Ratio of GMCs = 1.11, 95% CI 2-sided [0.88 to 1.4]
Statistical Analysis 10: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); HIb (Post-vaccination GMC; group ratio LA1:LA2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 1]; ANOVA; Ratio of GMCs = 1.27, 95% CI 2-sided [0.98 to 1.65]
Statistical Analysis 11: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); PnC 4 (Post-vaccination GMC; group ratio LA1:LA2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 1]; ANOVA; Ratio of GMCs = 0.92, 95% CI 2-sided [0.78 to 1.09]
Statistical Analysis 12: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); PnC 6B (Post-vaccination GMC; group ratio LA1:LA2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 1]; ANOVA; Ratio of GMCs = 0.97, 95% CI 2-sided [0.74 to 1.27]
Statistical Analysis 13: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); PnC 9V (Post-vaccination GMC; group ratio LA1:LA2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 1]; ANOVA; Ratio of GMCs = 0.86, 95% CI 2-sided [0.71 to 1.04]
Statistical Analysis 14: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); PnC 14 (Post-vaccination GMC; group ratio LA1:LA2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 1]; ANOVA; Ratio of GMCs = 0.91, 95% CI 2-sided [0.72 to 1.14]
Statistical Analysis 15: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); PnC 18C (Post-vaccination GMC; group ratio LA1:LA2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 1]; ANOVA; Ratio of GMCs = 0.89, 95% CI 2-sided [0.74 to 1.08]
Statistical Analysis 16: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); PnC 19F (Post-vaccination GMC; group ratio LA1:LA2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 1]; ANOVA; Ratio of GMCs = 0.9, 95% CI 2-sided [0.74 to 1.1]
Statistical Analysis 17: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); PnC 23F (Post-vaccination GMC; group ratio LA1:LA2); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 1]; ANOVA; Ratio of GMCs = 0.77, 95% CI 2-sided [0.6 to 0.99]
Statistical Analysis 18: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); Diphtheria (Post-vaccination GMC; group ratio LA3:LA4); Test type: Non-Inferiority or Equivalence — To assess non-inferiority of LA3 over LA4, the lower limit of two-sided 95% CI for the ratio of pertussis GMCs (GMCLA3 / GMCLA4) must be greater than 0.67; the lower limit of the two-sided 95% CI for the ratio of GMCs (GMCLA3 / GMCLA4) or GMTs (poliovirus antigens) for the other antigens must be greater than 0.50; ANOVA; Ratio of GMCs = 0.82, 95% CI 2-sided [0.69 to 0.99]
Statistical Analysis 19: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); Tetanus (Post-vaccination GMC; group ratio LA3:LA4); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 18]; ANOVA; Ratio of GMCs = 0.95, 95% CI 2-sided [0.83 to 1.09]
Statistical Analysis 20: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); PT (Post-vaccination GMC; group ratio LA3:LA4); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 18]; ANOVA; Ratio of GMCs = 0.93, 95% CI [0.78 to 1.1]
Statistical Analysis 21: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); FHA (Post-vaccination GMC; group ratio LA3:LA4); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 18]; ANOVA; Ratio of GMCs = 0.88, 95% CI 2-sided [0.75 to 1.03]
Statistical Analysis 22: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); Pertactin (Post-vaccination GMC; group ratio LA3:LA4; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 18]; ANOVA; Ratio of GMCs = 0.8, 95% CI 2-sided [0.66 to 0.97]
Statistical Analysis 23: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); Polio Type 1 (Post-vaccination GMT; group ratio LA3:LA4); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 18]; ANOVA; Ratio of GMTs = 0.78, 95% CI 2-sided [0.6 to 1.02]
Statistical Analysis 24: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); Polio Type 2 (Post-vaccination GMT; group ratio LA3:LA4); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 18]; ANOVA; Ratio of GMTs = 0.83, 95% CI 2-sided [0.63 to 1.09]
Statistical Analysis 25: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); Polio Type 3 (Post-vaccination GMT; group ratio LA3:LA4); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 18]; ANOVA; Ratio of GMTs = 0.81, 95% CI 2-sided [0.59 to 1.11]
Statistical Analysis 26: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); Hepatitis B (Post-vaccination GMT; group ratio LA3:LA4); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 18]; ANOVA; Ratio of GMTs = 0.95, 95% CI 2-sided [0.76 to 1.19]
Statistical Analysis 27: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); HIb (Post-vaccination GMC; group ratio LA3:LA4); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 18]; ANOVA; Ratio of GMCs = 1.07, 95% CI 2-sided [0.83 to 1.37]
Statistical Analysis 28: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); PnC 4 (Post-vaccination GMT; group ratio LA3:LA4); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 18]; ANOVA; Ratio of GMTs = 0.8, 95% CI 2-sided [0.68 to 0.95]
Statistical Analysis 29: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); PnC 6B (Post-vaccination GMC; group ratio LA3:LA4); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 18]; ANOVA; Ratio of GMCs = 0.87, 95% CI 2-sided [0.67 to 1.14]
Statistical Analysis 30: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); PnC 9V (Post-vaccination GMC; group ratio LA3:LA4); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 18]; ANOVA; Ratio of GMCs = 0.83, 95% CI 2-sided [0.69 to 1]
Statistical Analysis 31: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); PnC 14 (Post-vaccination GMC; group ratio LA3:LA4); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 18]; ANOVA; Ratio of GMCs = 0.84, 95% CI [0.67 to 1.05]
Statistical Analysis 32: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); PnC 18C (Post-vaccination GMC; group ratio LA3:LA4); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 18]; ANOVA; Ratio of GMCs = 0.75, 95% CI 2-sided [0.62 to 0.9]
Statistical Analysis 33: Comparison: LA4 (Infant Vaccines Only); PnC 19F (Post-vaccination GMC; group ratio LA3:LA4); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 18]; ANOVA; Ratio of GMCs = 0.91, 95% CI 2-sided [0.75 to 1.1]
Statistical Analysis 34: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); PnC 23F (Post-vaccination GMC; group ratio LA3:LA4); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 18]; ANOVA; Ratio of GMCs = 0.88, 95% CI 2-sided [0.69 to 1.12]

21. Secondary Outcome: Seroresponse Rates to DTaP, HBV, Hib, Pneumococcal and Polio Antigens at 1 Month After Infant Series Vaccination - LA Subjects
Description: as for outcome 19
Time Frame: 7 months of age (one month post-infant series)
Population: Per Protocol
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | LA1 (Men ACWY-CRM + Infant Vaccines) | LA2 (Infant Vaccines Only) | LA3 (Men ACWY-CRM + Infant Vaccines) | LA4 (Infant Vaccines Only)
Number analyzed (Participants) | 287 | 123 | 283 | 137
Percentages of subjects
  Diphtheria(≥ 0.1 IU/mL) (N=287,N=123,N=283,N=137) | 99 [96 to 100] | 98 [94 to 100] | 99 [96 to 100] | 99 [95 to 100]
  Tetanus (≥ 0.1 IU/mL) (N=287,N=123,N=283,N=137) | 100 [98 to 100] | 100 [97 to 100] | 100 [99 to 100] | 100 [97 to 100]
  PT(≥ 4-fold rise) (N=285,N=123, N=281,N=135) | 85 [81 to 89] | 86 [79 to 92] | 85 [80 to 89] | 82 [75 to 88]
  FHA (≥ 4-fold rise) (N=286,N=123, N=281,N=135) | 84 [79 to 88] | 86 [79 to 92] | 82 [77 to 86] | 81 [74 to 88]
  Pertactin(≥ 4-fold rise)(N=286,N=123,N=281,N=135) | 81 [76 to 85] | 87 [80 to 92] | 86 [82 to 90] | 88 [81 to 93]
  Polio Type 1 (≥1:8) (N=265,N=112,N=252,N=120) | 98 [95 to 99] | 100 [97 to 100] | 99 [97 to 100] | 98 [94 to 100]
  Polio Type 2 (≥1:8) (N=265,N=112,N=252,N=120) | 97 [95 to 99] | 99 [95 to 100] | 98 [95 to 99] | 98 [93 to 99]
  Polio Type 3 (≥1:8) (N=265,N=112,N=252,N=120) | 97 [95 to 99] | 97 [92 to 99] | 96 [93 to 98] | 97 [92 to 99]
  Hepatitis B(≥10 mIU/mL)(N=243,N=104,N=237,N=118) | 100 [98 to 100] | 100 [97 to 100] | 100 [98 to 100] | 100 [97 to 100]
  Hib (≥0.15 μg/mL) (N=287,N=123,N=283,N=137) | 99 [98 to 100] | 98 [94 to 100] | 97 [94 to 99] | 99 [96 to 100]
  Hib (≥1.0 μg/mL) (N=287,N=123,N=283,N=137) | 95 [92 to 97] | 93 [88 to 97] | 93 [90 to 96] | 96 [91 to 98]
  PnC 4 (≥ 0.35 μg/mL) (N=268,N=116,N=256,N=126) | 99 [96 to 100] | 99 [95 to 100] | 97 [94 to 99] | 98 [94 to 100]
  PnC 6B (≥ 0.35 μg/mL) (N=264,N=116,N=255,N=124) | 91 [86 to 94] | 86 [79 to 92] | 91 [87 to 95] | 90 [83 to 94]
  PnC 9V (≥ 0.35 μg/mL) (N=268,N=116,N=256,N=126) | 97 [95 to 99] | 98 [94 to 100] | 97 [94 to 99] | 96 [91 to 99]
  PnC 14 (≥ 0.35 μg/mL) (N=268,N=116,N=256,N=126) | 99 [97 to 100] | 97 [93 to 99] | 98 [95 to 99] | 98 [94 to 100]
  PnC 18C(≥ 0.35 μg/mL) (N=268,N=116,N=256, N=126) | 97 [94 to 98] | 98 [94 to 100] | 95 [91 to 97] | 98 [94 to 100]
  PnC 19F (≥ 0.35 μg/mL)(N=268,N=116,N=254,N=126) | 97 [94 to 98] | 98 [94 to 100] | 98 [96 to 100] | 96 [91 to 99]
  PnC 23F (≥ 0.35 μg/mL)(N=267,N=115,N=256, N=125) | 93 [89 to 96] | 97 [91 to 99] | 95 [91 to 97] | 94 [88 to 97]
Statistical Analysis 1: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); Diphtheria (Seroconversion percentage difference (PLA1 - PLA2)); Test type: Non-Inferiority or Equivalence — To assess non-inferiority of LA1 to LA2, the lower limit of the 95% CI for the difference in seroresponse rates (PLA1 - PLA2) must be greater than -5% for poliovirus and greater than -10% for all other antigens; ANOVA; Seroconversion Percentage difference = 0, 95% CI 2-sided [-2.2 to 4.4]
Statistical Analysis 2: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines); Tetanus (Seroconversion percentage difference (PLA1 - PLA2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 1]; ANOVA; Seroconversion Percentage difference = 0, 95% CI 2-sided [-1.9 to 2.6]
Statistical Analysis 3: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); PT (Seroconversion percentage difference (PLA1 - PLA2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 1]; ANOVA; Seroconversion Percentage difference = -1, 95% CI 2-sided [-7.7 to 7.1]
Statistical Analysis 4: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); FHA(Seroconversion percentage difference (PLA1 - PLA2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 1]; ANOVA; Seroconversion Percentage difference = -2, 95% CI 2-sided [-9.2 to 5.8]
Statistical Analysis 5: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); Pertactin (Seroconversion percentage difference (PLA1 - PLA2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 1]; ANOVA; Seroconversion Percentage difference = -6, 95% CI [-12.9 to 2.2]
Statistical Analysis 6: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); Polio Type 1 (Seroconversion percentage difference (PLA1 - PLA2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 1]; ANOVA; Seroconversion Percentage difference = -2, 95% CI 2-sided [-4.8 to 1.0]
Statistical Analysis 7: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); Polio Type 2 (Seroconversion percentage difference (PLA1 - PLA2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 1]; ANOVA; Seroconversion Percentage difference = -2, 95% CI 2-sided [-4.6 to 2.3]
Statistical Analysis 8: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); Polio Type 3 (Seroconversion percentage difference (PLA1 - PLA2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 1]; ANOVA; Seroconversion Percentage difference = 0, 95% CI 2-sided [-3.2 to 5.1]
Statistical Analysis 9: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); Hepatitis B (Seroconversion percentage difference (PLA1 - PLA2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 1]; ANOVA; Seroconversion Percentage difference = 0, 95% CI 2-sided [-1.5 to 3.5]
Statistical Analysis 10: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); Hib (≥ 0.15 μg/mL)(Seroconversion percentage difference (PLA1 - PLA2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 1]; ANOVA; Seroconversion Percentage difference = 1, 95% CI 2-sided [-1.1 to 5]
Statistical Analysis 11: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); Hib (≥1.0 μg/mL)(Seroconversion percentage difference (PLA1 - PLA2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 1]; ANOVA; Seroconversion Percentage difference = 2, 95% CI [-2.8 to 7.7]
Statistical Analysis 12: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); PnC 4(Seroconversion percentage difference (PLA1 - PLA2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 1]; ANOVA; Seroconversion Percentage difference = -1, 95% CI 2-sided [-3 to 3.3]
Statistical Analysis 13: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); PnC 6B(Seroconversion percentage difference (PLA1 - PLA2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 1]; ANOVA; Seroconversion Percentage difference = 4, 95% CI 2-sided [-2.2 to 12.3]
Statistical Analysis 14: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); PnC 9V (Seroconversion percentage difference (PLA1 - PLA2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 1]; ANOVA; Seroconversion Percentage difference = -1, 95% CI 2-sided [-3.9 to 3.6]
Statistical Analysis 15: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); PnC 14 (Seroconversion percentage difference (PLA1 - PLA2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 1]; ANOVA; Seroconversion Percentage difference = 1, 95% CI 2-sided [-1.1 to 6.2]
Statistical Analysis 16: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); PnC 18C (Seroconversion percentage difference (PLA1 - PLA2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 1]; ANOVA; Seroconversion Percentage difference = -2, 95% CI 2-sided [-4.8 to 2.9]
Statistical Analysis 17: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); PnC 19F (Seroconversion percentage difference (PLA1 - PLA2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 1]; ANOVA; Seroconversion Percentage difference = -2, 95% CI 2-sided [-4.8 to 2.9]
Statistical Analysis 18: Comparison: LA1 (Men ACWY-CRM + Infant Vaccines) vs LA2 (Infant Vaccines Only); PnC 23F (Seroconversion percentage difference (PLA1 - PLA2)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 1]; ANOVA; Seroconversion Percentage difference = -4, 95% CI 2-sided [-8 to 1.9]
Statistical Analysis 19: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); Diphtheria (Seroconversion percentage difference (PLA3 - PLA4)); Test type: Non-Inferiority or Equivalence — To assess non-inferiority of LA3 over LA4, the lower limit of the two-sided 95% CI for the difference in seroresponse rates (PLA3 - PLA4) must be greater than 5% for poliovirus and greater than -10% for all other antigens; ANOVA; Seroconversion Percentage difference = 0, 95% CI 2-sided [-2.3 to 3.8]
Statistical Analysis 20: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); Tetanus (Seroconversion percentage difference (PLA3 - PLA4)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 19]; ANOVA; Seroconversion Percentage difference = 0, 95% CI [-1.3 to 2.7]
Statistical Analysis 21: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); PT (Seroconversion percentage difference (PLA3 - PLA4)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 19]; Seroconversion Percentage difference; Seroconversion Percentage difference = 2, 95% CI 2-sided [-4.8 to 10.7]
Statistical Analysis 22: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); FHA(Seroconversion percentage difference (PLA3 - PLA4)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 19]; ANOVA; Seroconversion Percentage difference = 0, 95% CI 2-sided [-7.1 to 8.8]
Statistical Analysis 23: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); Pertactin (Seroconversion percentage difference (PLA3 - PLA4)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 19]; ANOVA; Seroconversion Percentage difference = -2, 95% CI 2-sided [-8 to 5.7]
Statistical Analysis 24: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); Polio Type 1 (Seroconversion percentage difference (PLA3 - PLA4)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 19]; ANOVA; Seroconversion Percentage difference = 0, 95% CI 2-sided [-2 to 4.7]
Statistical Analysis 25: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); Polio Type 2 (Seroconversion percentage difference (PLA3 - PLA4)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 19]; ANOVA; Seroconversion Percentage difference = 0, 95% CI 2-sided [-3 to 4.8]
Statistical Analysis 26: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); Polio Type 3 (Seroconversion percentage difference (PLA3 - PLA4)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 19]; ANOVA; Seroconversion Percentage difference = -1, 95% CI 2-sided [-4.4 to 4.5]
Statistical Analysis 27: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); Hepatitis B (Seroconversion percentage difference (PLA3 - PLA4)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 19]; ANOVA; Seroconversion Percentage difference = 0, 95% CI 2-sided [-2.3 to 2.7]
Statistical Analysis 28: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); Hib (≥ 0.15 μg/mL)(Seroconversion percentage difference (PLA3 - PLA4)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 19]; ANOVA; Seroconversion Percentage difference = -2, 95% CI 2-sided [-5.3 to 1]
Statistical Analysis 29: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); Hib (≥1.0 μg/mL)(Seroconversion percentage difference (PLA3 - PLA4)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 19]; ANOVA; Seroconversion Percentage difference = -2, 95% CI [-6.6 to 3]
Statistical Analysis 30: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); PnC 4 (Seroconversion percentage difference (PLA3 - PLA4)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 19]; ANOVA; Seroconversion Percentage difference = -1, 95% CI 2-sided [-4.2 to 3]
Statistical Analysis 31: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); PnC 6B (Seroconversion percentage difference (PLA3 - PLA4)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 19]; ANOVA; Seroconversion Percentage difference = 2, 95% CI 2-sided [-4 to 9]
Statistical Analysis 32: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); PnC 9V (Seroconversion percentage difference (PLA3 - PLA4)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 19]; ANOVA; Seroconversion Percentage difference = 1, 95% CI 2-sided [-2.8 to 6]
Statistical Analysis 33: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); PnC 14 (Seroconversion percentage difference (PLA3 - PLA4)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 19]; ANOVA; Seroconversion Percentage difference = -1, 95% CI 2-sided [-3.7 to 3.4]
Statistical Analysis 34: Comparison: LA4 (Infant Vaccines Only); PnC 18C (Seroconversion percentage difference (PLA3 - PLA4)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 19]; ANOVA; Seroconversion Percentage difference = -3, 95% CI 2-sided [-7.2 to 0.8]
Statistical Analysis 35: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); PnC 19F (Seroconversion percentage difference (PLA3 - PLA4)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 19]; ANOVA; Seroconversion Percentage difference = 2, 95% CI 2-sided [-0.8 to 7.5]
Statistical Analysis 36: Comparison: LA3 (Men ACWY-CRM + Infant Vaccines) vs LA4 (Infant Vaccines Only); PnC 23F (Seroconversion percentage difference (PLA3 - PLA4)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 21, analysis 19]; ANOVA; Seroconversion Percentage difference = 1, 95% CI [-3.7 to 7]

22. Secondary Outcome: Percentage of Subjects With Persistence Antibodies hSBA ≥1:4 at 12 Months of Age- US Subject
Description: Persistence of Antibodies as measured by the percentage of subjects with serum bactericidal activity using human complement (hSBA) ≥ 1:4, directed against N.meningitidis serogroups A, C, W and Y.
Time Frame: 12 Months of Age (one month pre-toddler vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | US1A (MenACWY- CRM + Infant Vaccines) | US2 (Infant Vaccine Only)
Number analyzed (Participants) | 84 | 74
Percentages of subjects
  A (84, 74) | 12 [6 to 21] | 3 [0 to 9]
  C (86, 73) | 53 [42 to 64] | 8 [3 to 17]
  W (85, 73) | 80 [70 to 88] | 4 [1 to 12]
  Y (84, 68) | 74 [63 to 83] | 1 [0 to 8]

23. Secondary Outcome: Percentage of Subjects With Persistence Antibodies hSBA ≥1:8 at 12 Months of Age- US Subject
Description: Persistence of Antibodies as measured by the percentage of subjects with serum bactericidal activity using human complement (hSBA) ≥ 1:8, directed against N.meningitidis serogroups A, C, W and Y.
Time Frame: 12 Months of Age (one month pre-toddler vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | US1A (MenACWY- CRM + Infant Vaccines) | US2 (Infant Vaccine Only)
Number analyzed (Participants) | 84 | 74
Percentages of subjects
  A (84, 74) | 10 [4 to 18] | 1 [0.034 to 7]
  C (86, 73) | 50 [39 to 61] | 7 [2 to 15]
  W (85, 73) | 71 [60 to 80] | 4 [1 to 12]
  Y (84, 68) | 61 [49 to 71] | 1 [0.037 to 8]

24. Secondary Outcome: Persistence Antibodies Geometric Mean Titers - US Subject
Description: Geometric Mean hSBA Titers directed against N. meningitides serogroups A, C, W and Y was measured at 12 Months of Age.
Time Frame: 12 Months of Age (one month pre-toddler vaccination)
Population: The analysis was done on per protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | US1A (MenACWY- CRM + Infant Vaccines ) | US2 (Infant Vaccine Only)
Number analyzed (Participants) | 84 | 74
Titers
  A (84, 74) | 2.51 [2.14 to 2.96] | 2.14 [1.8 to 2.54]
  C (86, 73) | 7.72 [5.9 to 10] | 2.26 [1.69 to 3.03]
  W (85, 73) | 14 [11 to 18] | 2.21 [1.69 to 2.9]
  Y (84, 68) | 11 [8.76 to 15] | 2.14 [1.6 to 2.86]

25. Secondary Outcome: Percentage of Subjects With Persistence Antibodies hSBA ≥1:4 at 12 or 16 Months of Age- LA Subject
Description: as for outcome 22
Time Frame: 12 or 16 Months of Age (one month pre-toddler vaccination)
Population: The analysis was done on per protocol population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- LA1 (Men ACWY-CRM + Infant Vaccines) (12m): LA infants received MenACWY at 2 and 6 months of age and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. Group LA1 was randomized into LA1A and LA 1B subgroups.
- LA2 (Infant Vaccines Only) (12m): LA infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. These infants received one dose of MenACWY concomitantly with pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and a second dose of MenACWY at 15 months of age.
- LA3 (Men ACWY-CRM + Infant Vaccines) (16m): LA infants received MenACWY at 2, 4 and 6 months of age; and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, pneumococcal conjugate vaccine, and rotavirus vaccine. Group LA3 was further randomized into LA3A and LA3B subgroups.
- LA4 (Infant Vaccines Only) (12m): LA infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, pneumococcal conjugate vaccine, and rotavirus vaccine at 2, 4 and 6 months of age. These infants received one dose of MenACWY concomitantly with pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months and a second dose of MenACWY along with DTaP and Hib vaccines at 15 months of age.
Arm/Group | LA1 (Men ACWY-CRM + Infant Vaccines) (12m) | LA2 (Infant Vaccines Only) (12m) | LA3 (Men ACWY-CRM + Infant Vaccines) (16m) | LA4 (Infant Vaccines Only) (12m)
Number analyzed (Participants) | 206 | 78 | 229 | 102
Percentages of subjects
  A (205, 78, 229, 101) | 29 [23 to 36] | 1 [0.032 to 7] | 18 [14 to 24] | 1 [0.025 to 5]
  C (206, 78, 229, 102) | 62 [55 to 68] | 4 [1 to 11] | 32 [26 to 38] | 2 [0 to 7]
  W (198, 70, 218, 98) | 95 [92 to 98] | 4 [1 to 12] | 72 [66 to 78] | 5 [2 to 12]
  Y (195, 71, 212, 95) | 82 [76 to 87] | 3 [0 to 10] | 65 [58 to 71] | 2 [0 to 7]

26. Secondary Outcome: Percentage of Subjects With Persistence Antibodies hSBA ≥1:8 at 12 or 16 Months of Age- LA Subject
Description: as for outcome 23
Time Frame: 12 or 16 Months of Age (one month pre-toddler vaccination)
Population: The analysis was done on per protocol population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | LA1 (Men ACWY-CRM + Infant Vaccines) (12m) | LA2 (Infant Vaccines Only) (12m) | LA3 (Men ACWY-CRM + Infant Vaccines) (16m) | LA4 (Infant Vaccines Only) (12m)
Number analyzed (Participants) | 206 | 78 | 229 | 102
Percentages of subjects
  A (205, 78, 229, 101) | 25 [20 to 32] | 0 [0 to 5] | 15 [11 to 20] | 0 [0 to 4]
  C (206, 78, 229, 102) | 57 [50 to 64] | 4 [1 to 11] | 26 [20 to 32] | 1 [0.025 to 5]
  W (198, 70, 218, 98) | 85 [79 to 90] | 4 [1 to 12] | 63 [56 to 69] | 5 [2 to 12]
  Y (195, 71, 212, 95) | 72 [65 to 78] | 3 [0 to 10] | 52 [45 to 59] | 0 [0 to 4]

27. Secondary Outcome: Persistence Antibodies Geometric Mean Titers - LA Subjects
Description: Geometric Mean hSBA Titers directed against N. meningitidis serogroups A, C, W and Y was measured at 12 or 16 Months of Age.
Time Frame: 12 or 16 Months of Age (one month pre-toddler vaccination)
Population: The analysis was done on per protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | LA1 (Men ACWY-CRM + Infant Vaccines) (12m) | LA2 (Infant Vaccines Only) (12m) | LA3 (Men ACWY-CRM + Infant Vaccines) (16m) | LA4 (Infant Vaccines Only) (12m)
Number analyzed (Participants) | 206 | 78 | 229 | 102
Titers
  A (205, 78, 229, 101) | 4.26 [3.55 to 5.11] | 2.02 [1.7 to 2.4] | 2.96 [2.63 to 3.33] | 2.02 [1.74 to 2.35]
  C (206, 78, 229, 102) | 12 [9.33 to 15] | 2.18 [1.73 to 2.74] | 4.14 [3.54 to 4.84] | 2.05 [1.68 to 2.51]
  W (198, 70, 218, 98) | 31 [26 to 37] | 2.34 [1.79 to 3.05] | 14 [12 to 18] | 2.33 [1.86 to 2.91]
  Y (195, 71, 212, 95) | 18 [15 to 22] | 2.2 [1.7 to 2.84] | 9.45 [7.81 to 11] | 2.04 [1.64 to 2.55]

28. Secondary Outcome: Percentage of Subjects (95% CI) With hSBA ≥ 1:4 at 1 Month After Toddler MenACWY Vaccination - US Subjects
Description: Immunogenicity as measured by the percentage of subjects with serum bactericidal activity using human complement (hSBA) ≥ 1:4 , directed against N.meningitidis serogroups A, C, W and Y.
Time Frame: 13 months of age (one month post-toddler vaccination)
Population: The analysis was done on per protocol population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | US1A (MenACWY- CRM + Infant Vaccines ) | US2 (Infant Vaccine Only)
Number analyzed (Participants) | 84 | 74
Percentages of subjects
  A Pre-vaccination (84, 74) | 12 [6 to 21] | 3 [0 to 9]
  A Post-vaccination (84, 74) | 94 [87 to 98] | 78 [67 to 87]
  C Pre-vaccination (86, 73) | 53 [42 to 64] | 8 [3 to 17]
  C Post-vaccination (86, 73) | 99 [94 to 100] | 95 [87 to 98]
  W Pre-vaccination (85, 73) | 80 [70 to 88] | 4 [1 to 12]
  W Post-vaccination (85, 73) | 100 [6 to 100] | 73 [61 to 82]
  Y Pre-vaccination (84, 68) | 74 [63 to 83] | 1 [0.037 to 8]
  Y Post-vaccination (84, 68) | 100 [96 to 100] | 62 [49 to 73]

29. Secondary Outcome: Percentage of Subjects (95% CI) With hSBA ≥ 1:8 at 1 Month After Toddler MenACWY Vaccination - US Subjects
Description: Immunogenicity as measured by the percentage of subjects with serum bactericidal activity using human complement (hSBA) ≥ 1:8 , directed against N.meningitidis serogroups A, C, W and Y.
Time Frame: 13 months of age (one month post-toddler vaccination)
Population: The analysis was done on per protocol population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | US1A (MenACWY- CRM + Infant Vaccines ) | US2 (Infant Vaccine Only)
Number analyzed (Participants) | 84 | 74
Percentages of subjects
  A Pre-vaccination (84, 74) | 10 [4 to 18] | 1 [0.034 to 7]
  A Post-vaccination (84, 74) | 94 [87 to 98] | 72 [60 to 81]
  C Pre-vaccination (86, 73) | 50 [39 to 61] | 7 [2 to 15]
  C Post-vaccination (86, 73) | 98 [92 to 100] | 90 [81 to 96]
  W Pre-vaccination (85, 73) | 71 [60 to 80] | 4 [1 to 12]
  W Post-vaccination (85, 73) | 100 [96 to 100] | 58 [45 to 69]
  Y Pre-vaccination (84, 68) | 61 [49 to 71] | 1 [0.037 to 8]
  Y Post-vaccination (84, 68) | 100 [96 to 100] | 56 [43 to 68]

30. Secondary Outcome: Percentage of Subjects (95% CI) With hSBA ≥ 1:16 at 1 Month After Toddler MenACWY Vaccination - US Subjects
Description: Immunogenicity as measured by the percentage of subjects with serum bactericidal activity using human complement (hSBA) ≥ 1:16 , directed against N.meningitidis serogroups A, C, W and Y.
Time Frame: 13 months of age (one month post-toddler vaccination)
Population: The analysis was done on per protocol population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | US1A (MenACWY- CRM + Infant Vaccines ) | US2 (Infant Vaccine Only)
Number analyzed (Participants) | 86 | 74
Percentages of subjects
  A Pre-vaccination (84, 74) | 5 [1 to 12] | 1 [0.034 to 7]
  A Post-vaccination (84, 74) | 90 [82 to 96] | 55 [43 to 67]
  C Pre-vaccination (86, 73) | 35 [25 to 46] | 0 [0 to 5]
  C Post-vaccination (86, 73) | 95 [89 to 99] | 78 [67 to 87]
  W Pre-vaccination (85, 73) | 48 [37 to 59] | 3 [0 to 10]
  W Post-vaccination (85, 73) | 100 [96 to 100] | 38 [27 to 50]
  Y Pre-vaccination (84, 68) | 45 [34 to 56] | 1 [0.037 to 8]
  Y Post-vaccination (84, 68) | 100 [96 to 100] | 41 [29 to 54]

31. Secondary Outcome: Geometric Mean hSBA Titers at 1 Month After Toddler MenACWY Vaccination - US Subjects
Description: as for outcome 4
Time Frame: 13 months of age (one month post-toddler vaccination)
Population: The analysis was done on per protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | US1A (MenACWY- CRM + Infant Vaccines ) | US2 (Infant Vaccine Only)
Number analyzed (Participants) | 84 | 74
Titers
  A Pre-vaccination (84, 74) | 2.51 [2.14 to 2.96] | 2.14 [1.8 to 2.54]
  A Post-vaccination (84, 74) | 77 [55 to 109] | 17 [12 to 25]
  C Pre-vaccination (86, 73) | 7.72 [5.9 to 10] | 2.26 [1.69 to 3.03]
  C Post-vaccination (86, 73) | 227 [155 to 332] | 35 [23 to 54]
  W Pre-vaccination (85, 73) | 14 [11 to 18] | 2.21 [1.69 to 2.9]
  W Post-vaccination (85, 73) | 416 [288 to 602] | 11 [7.59 to 17]
  Y Pre-vaccination (84, 68) | 11 [8.76 to 15] | 2.14 [1.6 to 2.86]
  Y Post-vaccination (84, 68) | 395 [269 to 580] | 10 [6.72 to 16]

32. Secondary Outcome: Percentage of Subjects (95% CI) With hSBA ≥1:4 at 1 Month After Toddler MenACWY Vaccination - LA Subjects
Description: Immunogenicity as measured by the percentage of subjects with serum bactericidal activity using human complement (hSBA) ≥ 1:4, directed against N. meningitidis serogroups A, C, W and Y.
Time Frame: 13 or 17 Months of Age (one month post-toddler vaccination)
Population: The analysis was done on per protocol population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- LA1A (Men ACWY-CRM + Infant Vaccines): LA infants received MenACWY at 2 and 6 months of age; and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. These subjects received a third dose of MenACWY concomitantly with pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months of age.
- LA3A (Men ACWY-CRM + Infant Vaccines): LA infants received MenACWY at 2, 4 and 6 months of age; and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, pneumococcal conjugate vaccine, and rotavirus vaccine. Around 12 months of age, these infants were recommended to receive pneumococcal conjugate vaccine, HAV, and MMR-V. At 16 months of age, these subjects received the fourth dose of MenACWY along with concomitant DTaP and Hib.
Arm/Group | LA1A (Men ACWY-CRM + Infant Vaccines) | LA3A (Men ACWY-CRM + Infant Vaccines)
Number analyzed (Participants) | 103 | 122
Percentages of subjects
  A Pre-vaccination (103, 120) | 28 [20 to 38] | 18 [12 to 26]
  A Post-vaccination (103,120) | 94 [88 to 98] | 95 [89 to 98]
  C Pre-vaccination (102,122) | 61 [51 to 70] | 30 [22 to 38]
  C Post-vaccination (102,122) | 98 [93 to 100] | 98 [94 to 100]
  W Pre-vaccination (98,112) | 97 [91 to 99] | 71 [61 to 79]
  W Post-vaccination (98,112) | 100 [96 to 100] | 100 [97 to 100]
  Y Pre-vaccination (98,109) | 78 [68 to 85] | 61 [52 to 71]
  Y Post-vaccination (98,109) | 99 [94 to 100] | 99 [95 to 100]

33. Secondary Outcome: Percentage of Subjects (95% CI) With hSBA ≥1:8 at 1 Month After Toddler MenACWY Vaccination - LA Subjects
Description: Immunogenicity as measured by the percentage of subjects with serum bactericidal activity using human complement (hSBA) ≥ 1:8, directed against N. meningitidis serogroups A, C, W and Y.
Time Frame: 13 or 17 Months of Age (one month post-toddler vaccination)
Population: The analysis was done on per protocol population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | LA1A (Men ACWY-CRM + Infant Vaccines) | LA3A (Men ACWY-CRM + Infant Vaccines)
Number analyzed (Participants) | 103 | 122
Percentages of subjects
  A Pre-vaccination (103, 120) | 23 [16 to 33] | 13 [8 to 21]
  A Post-vaccination (103,120) | 94 [88 to 98] | 95 [89 to 98]
  C Pre-vaccination (102,122) | 57 [47 to 67] | 22 [15 to 31]
  C Post-vaccination (102,122) | 97 [92 to 99] | 98 [94 to 100]
  W Pre-vaccination (98,112) | 84 [75 to 90] | 62 [52 to 71]
  W Post-vaccination (98,112) | 99 [94 to 100] | 100 [97 to 100]
  Y Pre-vaccination (98,109) | 67 [57 to 76] | 47 [37 to 57]
  Y Post-vaccination (98,109) | 99 [94 to 100] | 99 [95 to 100]

34. Secondary Outcome: Percentage of Subjects With hSBA ≥ 1:16 at 1 Month After Toddler MenACWY Vaccination - LA Subjects
Description: Immunogenicity as measured by the percentage of subjects with serum bactericidal activity using human complement (hSBA) ≥ 1:16, directed against N. meningitidis serogroups A, C, W and Y.
Time Frame: 13 or 17 Months of Age (one month post-toddler vaccination)
Population: The analysis was done on per protocol population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | LA1A (Men ACWY-CRM + Infant Vaccines) | LA3A (Men ACWY-CRM + Infant Vaccines)
Number analyzed (Participants) | 103 | 122
Percentages of subjects
  A Pre-vaccination (103, 120) | 16 [9 to 24] | 9 [5 to 16]
  A Post-vaccination (103, 120) | 93 [86 to 97] | 94 [88 to 98]
  C Pre-vaccination (102, 122) | 47 [37 to 57] | 18 [12 to 26]
  C Post-vaccination (102, 122) | 95 [89 to 98] | 96 [91 to 99]
  W Pre-vaccination (98,112) | 64 [54 to 74] | 50 [40 to 60]
  W Post-vaccination (98, 112) | 99 [94 to 100] | 100 [97 to 100]
  Y Pre-vaccination (98,109) | 53 [43 to 63] | 32 [23 to 42]
  Y Post-vaccination (98, 109) | 99 [94 to 100] | 98 [94 to 100]

35. Secondary Outcome: Geometric Mean hSBA Titers at 1 Month After Toddler MenACWY Vaccination - LA Subjects
Description: Immunogenicity as measured by Serum bactericidal activity using human complement (hSBA) GMTs, directed against N. meningitidis serogroups A, C, W and Y.
Time Frame: 13 or 17 Months of Age (one month post-toddler vaccination)
Population: The analysis was done on per protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | LA1A (Men ACWY-CRM + Infant Vaccines) | LA3A (Men ACWY-CRM + Infant Vaccines)
Number analyzed (Participants) | 103 | 122
Titers
  A Pre-vaccination (103, 120) | 3.83 [3.3 to 4.45] | 2.95 [2.57 to 3.39]
  A Post-vaccination (103, 120) | 112 [85 to 148] | 146 [113 to 188]
  C Pre-vaccination (102, 122) | 11 [8.91 to 13] | 3.83 [3.2 to 4.6]
  C Post-vaccination (102, 122) | 279 [218 to 358] | 283 [225 to 355]
  W Pre-vaccination (98, 112) | 28 [22 to 34] | 13 [11 to 16]
  W Post-vaccination (98, 112) | 762 [604 to 960] | 727 [586 to 903]
  Y Pre-vaccination (98, 109) | 16 [13 to 20] | 8.1 [6.58 to 9.96]
  Y Post-vaccination (98, 109) | 550 [426 to 710] | 590 [463 to 751]

36. Secondary Outcome: Geometric Mean Concentrations of Pneumococcal Antibodies at 1 Month After Toddler Vaccination - US Subjects
Description: Immunogenicity as measured by antibody GMTs, directed against pneumococcal antigens PnC 4, PnC 6B, PnC 9V, PnC 14, PnC 18C, PnC 19F and PnC 23F.
Time Frame: 13 months of age (one month post-toddler vaccination)
Population: Per Protocol
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | US1A (MenACWY-CRM + Infant Vaccines) | US1B (MenACWY-CRM + Infant Vaccines)
Number analyzed (Participants) | 87 | 99
Titers
  PnC 4 (N=86, N=99) | 2.9 [2.33 to 3.61] | 3.24 [2.64 to 3.97]
  PnC 6B (N=86, N=99) | 6.82 [5.67 to 8.21] | 8.58 [7.22 to 10]
  PnC 9V (N=86, N=99) | 2.8 [2.26 to 3.47] | 3.13 [2.56 to 3.82]
  PnC 14 (N=86, N=99) | 12 [9.74 to 14] | 15 [12 to 17]
  PnC 18C (N=87, N=98) | 2.76 [2.26 to 3.38] | 2.71 [2.24 to 3.27]
  PnC 19F(N=86, N=99) | 3.63 [3 to 4.39] | 3.48 [2.92 to 4.16]
  PnC 23F (N=87, N=99) | 5.31 [4.2 to 6.71] | 5.63 [4.52 to 7.01]
Statistical Analysis 1: Comparison: US1A (MenACWY-CRM + Infant Vaccines) vs US1B (MenACWY-CRM + Infant Vaccines); PnC 4 (Post-vaccination GMC; group ratio US1A:US1B); Test type: Non-Inferiority or Equivalence — To assess non-inferiority of US1A over US1B, the lower limit of 95% CI for the ratio of pneumococcal GMCs (GMCUS1A / GMCUS1B) had to be greater than 0.50; ANOVA; Ratio of GMCs = 0.9, 95% CI 2-sided [0.67 to 1.2]
Statistical Analysis 2: Comparison: US1A (MenACWY-CRM + Infant Vaccines) vs US1B (MenACWY-CRM + Infant Vaccines); PnC 6B (Post-vaccination GMC; group ratio US1A:US1B); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 36, analysis 1]; ANOVA; Ratio of GMCs = 0.8, 95% CI 2-sided [0.62 to 1.02]
Statistical Analysis 3: Comparison: US1A (MenACWY-CRM + Infant Vaccines) vs US1B (MenACWY-CRM + Infant Vaccines); PnC 9V (Post-vaccination GMC; group ratio US1A:US1B); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 36, analysis 1]; ANOVA; Ratio of GMCs = 0.89, 95% CI 2-sided [0.67 to 1.2]
Statistical Analysis 4: Comparison: US1A (MenACWY-CRM + Infant Vaccines) vs US1B (MenACWY-CRM + Infant Vaccines); PnC 14 (Post-vaccination GMC; group ratio US1A:US1B); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 36, analysis 1]; ANOVA; Ratio of GMCs = 0.8, 95% CI 2-sided [0.63 to 1.03]
Statistical Analysis 5: Comparison: US1A (MenACWY-CRM + Infant Vaccines) vs US1B (MenACWY-CRM + Infant Vaccines); PnC 18C (Post-vaccination GMC; group ratio US1A:US1B); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 36, analysis 1]; ANOVA; Ratio of GMCs = 1.02, 95% CI 2-sided [0.78 to 1.34]
Statistical Analysis 6: Comparison: US1A (MenACWY-CRM + Infant Vaccines) vs US1B (MenACWY-CRM + Infant Vaccines); PnC 19F (Post-vaccination GMC; group ratio US1A:US1B); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 36, analysis 1]; ANOVA; Ratio of GMCs = 1.04, 95% CI [0.81 to 1.34]
Statistical Analysis 7: Comparison: US1A (MenACWY-CRM + Infant Vaccines) vs US1B (MenACWY-CRM + Infant Vaccines); PnC 23F (Post-vaccination GMC; group ratio US1A:US1B); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 36, analysis 1]; ANOVA; Ratio of GMCs = 0.94, 95% CI 2-sided [0.69 to 1.29]

37. Secondary Outcome: Percentage of Subjects With Pneumococcal Antibody GMCs ≥1.0 μg/mL at 1 Month After Toddler Vaccination - US Subjects
Description: Immunogenicity as measured by Percentage of Subjects with Pneumococcal Antibody GMCs ≥1.0 μg/mL directed against pneumococcal antigens PnC 4, PnC 6B, PnC 9V, PnC 14, PnC 18C, PnC 19F and PnC 23F.
Time Frame: 13 months of age (one month post-toddler vaccination)
Population: Per Protocol
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | US1A (MenACWY-CRM + Infant Vaccines) | US1B (MenACWY-CRM + Infant Vaccines) | US2 (Infant Vaccines Only)
Number analyzed (Participants) | 87 | 99 | 81
Percentages of subjects
  PnC 4 (N=86, N=99, N=81) | 91 [82 to 96] | 90 [82 to 95] | 84 [74 to 91]
  PnC 6B (N=86, N=99, N=80) | 100 [96 to 100] | 96 [90 to 99] | 99 [93 to 100]
  PnC 9V (N=86, N=99, N=80) | 87 [78 to 93] | 91 [83 to 96] | 86 [77 to 93]
  PnC 14 (N=86, N=99, N=81) | 99 [94 to 100] | 100 [96 to 100] | 100 [96 to 100]
  PnC 18C (N=87, N=98, N=81) | 86 [77 to 93] | 92 [85 to 96] | 94 [86 to 98]
  PnC 19F(N=86, N=99, N=80) | 97 [90 to 99] | 93 [86 to 97] | 99 [93 to 100]
  PnC 23F (N=87, N=99, N=80) | 93 [86 to 97] | 95 [89 to 98] | 99 [93 to 100]
Statistical Analysis 1: Comparison: US1A (MenACWY-CRM + Infant Vaccines) vs US1B (MenACWY-CRM + Infant Vaccines); PnC 4 (percentage difference (US1A - US1B)); Test type: Non-Inferiority or Equivalence — To assess non-inferiority of US1A over US1B, the lower limit of 95% CI for the difference in rates (PUS1A - PUS1B) had to be greater than -10%; ANOVA; Percentage difference = 1, 95% CI 2-sided [-8 to 10]
Statistical Analysis 2: Comparison: US1A (MenACWY-CRM + Infant Vaccines) vs US1B (MenACWY-CRM + Infant Vaccines); PnC 6B (percentage difference (US1A - US1B)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 37, analysis 1]; ANOVA; Percentage difference = 4, 95% CI 2-sided [0 to 10]
Statistical Analysis 3: Comparison: US1A (MenACWY-CRM + Infant Vaccines) vs US1B (MenACWY-CRM + Infant Vaccines); PnC 9V (percentage difference (US1A - US1B)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 37, analysis 1]; ANOVA; Percentage difference = -4, 95% CI 2-sided [-13 to 5]
Statistical Analysis 4: Comparison: US1A (MenACWY-CRM + Infant Vaccines) vs US1B (MenACWY-CRM + Infant Vaccines); PnC 14 (percentage difference (US1A - US1B)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 37, analysis 1]; ANOVA; Percentage difference = -1, 95% CI 2-sided [-6 to 3]
Statistical Analysis 5: Comparison: US1A (MenACWY-CRM + Infant Vaccines) vs US1B (MenACWY-CRM + Infant Vaccines); PnC 18C (percentage difference (US1A:US1B)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 37, analysis 1]; ANOVA; Percentage difference = -6, 95% CI 2-sided [-15 to 3]
Statistical Analysis 6: Comparison: US1A (MenACWY-CRM + Infant Vaccines) vs US1B (MenACWY-CRM + Infant Vaccines); PnC 19F (percentage difference (US1A:US1B)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 37, analysis 1]; ANOVA; Percentage difference = 4, 95% CI 2-sided [-4 to 11]
Statistical Analysis 7: Comparison: US1A (MenACWY-CRM + Infant Vaccines) vs US1B (MenACWY-CRM + Infant Vaccines); PnC 239F (percentage difference (US1A:US1B)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 37, analysis 1]; ANOVA; Percentage difference = -2, 95% CI 2-sided [-10 to 5]

38. Secondary Outcome: Geometric Mean Concentrations of Pneumococcal Antibodies at 1 Month After Toddler Vaccination - LA Subjects
Description: as for outcome 36
Time Frame: 13 months of age (one month post-toddler vaccination)
Population: Per Protocol
Measure: Geometric Mean (95% Confidence Interval); unit: Concentrations (μg/mL)
Groups:
- LA1B (Men ACWY-CRM + Infant Vaccines): LA infants received MenACWY at 2 and 6 months of age and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. These subjects received pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months and a third dose of MenACWY at 13 months of age.
Arm/Group | LA1A (Men ACWY-CRM + Infant Vaccines) | LA1B (Men ACWY-CRM + Infant Vaccines)
Number analyzed (Participants) | 97 | 97
Concentrations (μg/mL)
  PnC 4 (N=97, N=97) | 3.16 [2.63 to 3.8] | 4.02 [3.34 to 4.83]
  PnC 6B (N=96, N=97) | 4.52 [3.42 to 5.97] | 5.61 [4.25 to 7.4]
  PnC 9V (N=97, N=97) | 2.79 [2.34 to 3.31] | 3.77 [3.17 to 4.48]
  PnC 14(N=97, N=97) | 8.91 [7.52 to 11] | 14 [12 to 16]
  PnC 18C (N=97, N=97) | 2.15 [1.79 to 2.58] | 2.77 [2.31 to 3.32]
  PnC 19F (N=97, N=97) | 3.26 [2.62 to 4.05] | 4.26 [3.43 to 5.29]
  PnC 23F (N=97, N=97) | 4.38 [3.51 to 5.48] | 5.92 [4.74 to 7.4]
Statistical Analysis 1: Comparison: LA1A (Men ACWY-CRM + Infant Vaccines) vs LA1B (Men ACWY-CRM + Infant Vaccines); PnC 4 (Post-vaccination GMC; group ratio LA1A:LA1B); Test type: Non-Inferiority or Equivalence — To assess non-inferiority of LA1A over LA1B, the lower limit of the two-sided 95% CI for the ratio of pneumococcal GMCs (GMCLA1A / GMCLA1B) had to be greater than 0.50; ANOVA; Ratio of GMCs = 0.79, 95% CI 2-sided [0.61 to 1.02]
Statistical Analysis 2: Comparison: LA1A (Men ACWY-CRM + Infant Vaccines) vs LA1B (Men ACWY-CRM + Infant Vaccines); PnC 6B (Post-vaccination GMC; group ratio LA1A:LA1B); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 38, analysis 1]; ANOVA; Ratio of GMCs = 0.81, 95% CI 2-sided [0.54 to 1.2]
Statistical Analysis 3: Comparison: LA1A (Men ACWY-CRM + Infant Vaccines) vs LA1B (Men ACWY-CRM + Infant Vaccines); PnC 9V (Post-vaccination GMC; group ratio LA1A:LA1B); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 38, analysis 1]; ANOVA; Ratio of GMCs = 0.74, 95% CI 2-sided [0.58 to 0.94]
Statistical Analysis 4: Comparison: LA1A (Men ACWY-CRM + Infant Vaccines) vs LA1B (Men ACWY-CRM + Infant Vaccines); PnC 14 (Post-vaccination GMC; group ratio LA1A:LA1B); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 38, analysis 1]; ANOVA; Ratio of GMCs = 0.65, 95% CI 2-sided [0.51 to 0.82]
Statistical Analysis 5: Comparison: LA1A (Men ACWY-CRM + Infant Vaccines) vs LA1B (Men ACWY-CRM + Infant Vaccines); PnC 18C (Post-vaccination GMC; group ratio LA1A:LA1B); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 38, analysis 1]; ANOVA; Ratio of GMCs = 0.78, 95% CI 2-sided [0.6 to 1.01]
Statistical Analysis 6: Comparison: LA1A (Men ACWY-CRM + Infant Vaccines) vs LA1B (Men ACWY-CRM + Infant Vaccines); PnC 19F (Post-vaccination GMC; group ratio LA1A:LA1B); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 38, analysis 1]; ANOVA; Ratio of GMCs = 0.77, 95% CI 2-sided [0.56 to 1.04]
Statistical Analysis 7: Comparison: LA1A (Men ACWY-CRM + Infant Vaccines) vs LA1B (Men ACWY-CRM + Infant Vaccines); PnC 23F (Post-vaccination GMC; group ratio LA1A:LA1B); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 38, analysis 1]; ANOVA; Ratio of GMCs = 0.74, 95% CI 2-sided [0.54 to 1.01]

39. Secondary Outcome: Percentage of Subjects With Pneumococcal Antibody Concentration ≥1.0 μg/mL at 1 Month After Toddler Vaccination - LA Subjects
Description: as for outcome 37
Time Frame: 13 months of age (one month post-toddler vaccination)
Population: Per Protocol
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | LA1A (Men ACWY-CRM + Infant Vaccines) | LA1B (Men ACWY-CRM + Infant Vaccines)
Number analyzed (Participants) | 97 | 97
Percentages of subjects
  PnC 4 (N=97, N=97) | 93 [86 to 97] | 95 [88 to 98]
  PnC 6B (N=96, N=97) | 86 [78 to 93] | 89 [81 to 94]
  PnC 9V (N=97, N=97) | 92 [84 to 96] | 95 [88 to 98]
  PnC 14 (N=97, N=97) | 99 [94 to 100] | 100 [96 to 100]
  PnC 18C (N=97, N=97) | 80 [71 to 88] | 95 [88 to 98]
  PnC 19F (N=97, N=97) | 90 [82 to 95] | 93 [86 to 97]
  PnC 23F (N=97, N=97) | 95 [88 to 98] | 95 [88 to 98]
Statistical Analysis 1: Comparison: LA1A (Men ACWY-CRM + Infant Vaccines) vs LA1B (Men ACWY-CRM + Infant Vaccines); PnC 4 (percentage difference (LA1A - LA1B)); Test type: Non-Inferiority or Equivalence — To assess non-inferiority of LA1A over LA1B, the lower limit of the two-sided 95% CI for the difference in rates (PLA1A - PLA1B) had to be greater than -10%; ANOVA; Percentage difference = -2, 95% CI 2-sided [-9.6 to 5.2]
Statistical Analysis 2: Comparison: LA1A (Men ACWY-CRM + Infant Vaccines) vs LA1B (Men ACWY-CRM + Infant Vaccines); PnC 6B (percentage difference (LA1A - LA1B)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 39, analysis 1]; ANOVA; Percentage difference = -2, 95% CI 2-sided [-11.9 to 7.3]
Statistical Analysis 3: Comparison: LA1A (Men ACWY-CRM + Infant Vaccines) vs LA1B (Men ACWY-CRM + Infant Vaccines); PnC 9V (percentage difference (LA1A - LA1B)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 39, analysis 1]; ANOVA; Percentage difference = -3, 95% CI 2-sided [-10.9 to 4.3]
Statistical Analysis 4: Comparison: LA1A (Men ACWY-CRM + Infant Vaccines) vs LA1B (Men ACWY-CRM + Infant Vaccines); PnC 14 (percentage difference (LA1A - LA1B)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 39, analysis 1]; ANOVA; Percentage difference = -1, 95% CI 2-sided [-5.6 to 2.7]
Statistical Analysis 5: Comparison: LA1A (Men ACWY-CRM + Infant Vaccines) vs LA1B (Men ACWY-CRM + Infant Vaccines); PnC 18C (percentage difference (LA1A - LA1B)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 39, analysis 1]; ANOVA; Percentage difference = -14, 95% CI 2-sided [-24.1 to -5.6]
Statistical Analysis 6: Comparison: LA1A (Men ACWY-CRM + Infant Vaccines) vs LA1B (Men ACWY-CRM + Infant Vaccines); PnC 19F (percentage difference (LA1A - LA1B)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 39, analysis 1]; ANOVA; Percentage difference = -3, 95% CI 2-sided [-11.6 to 5.2]
Statistical Analysis 7: Comparison: LA1A (Men ACWY-CRM + Infant Vaccines) vs LA1B (Men ACWY-CRM + Infant Vaccines); PnC 23F (percentage difference (LA1A - LA1B)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 39, analysis 1]; ANOVA; Percentage difference = 0, 95% CI 2-sided [-7 to 7]

40. Secondary Outcome: Geometric Mean Concentrations or Titers of DTaP and Hib Antigens at 1 Month After Toddler Vaccination - LA Subjects
Description: Immunogenicity as measured by antibody GMCs/GMTs, directed against DTaP and Hib Antigens
Time Frame: 17 months of age (one month post-toddler vaccination)
Population: Per Protocol
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- LA3B (Men ACWY-CRM + Infant Vaccines): LA infants received MenACWY at 2, 4 and 6 months of age; and as part of routine infant vaccination schedule received, DTaP-IPV-HBV, Hib, pneumococcal conjugate vaccine, and rotavirus vaccine. Around 12 months of age, received pneumococcal conjugate vaccine, HAV, and MMR-V. At 16 months of age, these subjects received DTaP and Hib. At 17 months of age, these subjects received the fourth dose of MenACWY.
Arm/Group | LA3A (Men ACWY-CRM + Infant Vaccines) | LA3B (Men ACWY-CRM + Infant Vaccines)
Number analyzed (Participants) | 118 | 101
Titers
  Diphtheria (N=118, N=101) | 5.4 [4.74 to 6.15] | 5.16 [4.48 to 5.94]
  Tetanus (N=118, N=101) | 6.17 [5.29 to 7.2] | 6.58 [5.57 to 7.77]
  PT (N=113, N=99) | 68 [58 to 80] | 62 [52 to 73]
  FHA (N=113, N=99) | 245 [208 to 288] | 215 [181 to 256]
  Pertactin (N=113, N=99) | 238 [198 to 286] | 197 [161 to 240]
  Hib (N=117, N=101) | 35 [28 to 43] | 41 [32 to 51]
Statistical Analysis 1: Comparison: LA3A (Men ACWY-CRM + Infant Vaccines) vs LA3B (Men ACWY-CRM + Infant Vaccines); Diphtheria (Post-vaccination GMC; group ratio LA3A:LA3B); Test type: Non-Inferiority or Equivalence — To assess non-inferiority of LA3A over LA3B, the lower limit of the two-sided 95% CI for the ratio of GMCs (GMCLA3A/GMCLA3B) had to be greater than 0.67 for PT, FHA and pertactin and greater than 0.50 for Hib, diphtheria and tetanus; ANOVA; Ratio of GMCs = 1.05, 95% CI 2-sided [0.86 to 1.27]
Statistical Analysis 2: Comparison: LA3A (Men ACWY-CRM + Infant Vaccines) vs LA3B (Men ACWY-CRM + Infant Vaccines); Tetanus (Post-vaccination GMC; group ratio LA3A:LA3B); Test type: Non-Inferiority or Equivalence — To assess non-inferiority of LA3A over LA3B, the lower limit of the two-sided 95% CI for the ratio of GMCs (GMCLA3A / GMCLA3B) had to be greater than 0.67 for PT, FHA and pertactin and greater than 0.50 for Hib, diphtheria and tetanus; ANOVA; Ratio of GMCs = 0.94, 95% CI 2-sided [0.75 to 1.18]
Statistical Analysis 3: Comparison: LA3A (Men ACWY-CRM + Infant Vaccines) vs LA3B (Men ACWY-CRM + Infant Vaccines); PT (Post-vaccination GMC; group ratio LA3A:LA3B); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 40, analysis 2]; ANOVA; Ratio of GMCs = 1.11, 95% CI 2-sided [0.88 to 1.4]
Statistical Analysis 4: Comparison: LA3A (Men ACWY-CRM + Infant Vaccines) vs LA3B (Men ACWY-CRM + Infant Vaccines); FHA (Post-vaccination GMC; group ratio LA3A:LA3B); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 40, analysis 2]; ANOVA; Ratio of GMCs = 1.14, 95% CI 2-sided [0.9 to 1.44]
Statistical Analysis 5: Comparison: LA3A (Men ACWY-CRM + Infant Vaccines) vs LA3B (Men ACWY-CRM + Infant Vaccines); Pertactin (Post-vaccination GMC; group ratio LA3A:LA3B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 40, analysis 2]; ANOVA; Ratio of GMCs = 1.21, 95% CI 2-sided [0.92 to 1.59]
Statistical Analysis 6: Comparison: LA3A (Men ACWY-CRM + Infant Vaccines) vs LA3B (Men ACWY-CRM + Infant Vaccines); Hib (Post-vaccination GMC; group ratio LA3A:LA3B); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 40, analysis 2]; ANOVA; Ratio of GMCs = 0.86, 95% CI 2-sided [0.63 to 1.16]

41. Secondary Outcome: Seroresponse Rates to DTaP and Hib Antigens at 1 Month After Toddler Vaccination - LA Subjects
Description: Immunogenicity as measured by Percentage of Subjects with predefined seroprotective antibody titers against DTaP and Hib Antigens
Time Frame: 17 months of age (one month post-toddler vaccination)
Population: Per Protocol
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | LA3A (Men ACWY-CRM + Infant Vaccines) | LA3B (Men ACWY-CRM + Infant Vaccines)
Number analyzed (Participants) | 118 | 101
Percentages of subjects
  Diphtheria (≥1.0 IU/mL) (N=118, N=101) | 98 [94 to 100] | 98 [93 to 100]
  Tetanus (≥1.0 IU/mL) (N=118, N=101) | 98 [94 to 100] | 98 [93 to 100]
  PT (≥4 fold rise) (N=113, N=99) | 89 [82 to 94] | 84 [75 to 90]
  FHA (≥4-fold rise) (N=113, N=99) | 87 [79 to 92] | 88 [80 to 94]
  Pertactin (≥4-fold rise) (N=113, N=99) | 89 [82 to 94] | 88 [80 to 94]
  Hib (≥0.15 μg/mL) (N=117, N=101) | 100 [97 to 100] | 100 [96 to 100]
  Hib (≥1.0 μg/mL) (N=117, N=101) | 100 [97 to 100] | 99 [95 to 100]
Statistical Analysis 1: Comparison: LA3A (Men ACWY-CRM + Infant Vaccines) vs LA3B (Men ACWY-CRM + Infant Vaccines); Diphtheria (percentage difference (LA3A - LA3B)); Test type: Non-Inferiority or Equivalence — To assess non-inferiority of LA3A over LA3B, The lower limit of the two-sided 95% CI for the difference (PLA3A-PLA3B) in percentages of subjects with seroresponse against diphtheria, tetanus, Hib and pertussis antigens (except FHA for ≥4 fold rise) was greater than -10%; ANOVA; Percentage difference = 0, 95% CI [-4.2 to 5.4]
Statistical Analysis 2: Comparison: LA3A (Men ACWY-CRM + Infant Vaccines) vs LA3B (Men ACWY-CRM + Infant Vaccines); Tetanus (percentage difference (LA3A - LA3B)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 41, analysis 1]; ANOVA; Percentage difference = 0, 95% CI 2-sided [-4.2 to 5.4]
Statistical Analysis 3: Comparison: LA3A (Men ACWY-CRM + Infant Vaccines) vs LA3B (Men ACWY-CRM + Infant Vaccines); PT (percentage difference (LA3A - LA3B)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 41, analysis 1]; ANOVA; Percentage difference = 6, 95% CI [-3.6 to 15.2]
Statistical Analysis 4: Comparison: LA3A (Men ACWY-CRM + Infant Vaccines) vs LA3B (Men ACWY-CRM + Infant Vaccines); FHA (percentage difference (LA3A - LA3B)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 41, analysis 1]; ANOVA; Percentage difference = -1, 95% CI 2-sided [-10.2 to 8.2]
Statistical Analysis 5: Comparison: LA3A (Men ACWY-CRM + Infant Vaccines) vs LA3B (Men ACWY-CRM + Infant Vaccines); Pertactin (percentage difference (LA3A - LA3B)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 41, analysis 1]; ANOVA; Percentage difference = 2, 95% CI 2-sided [-7.2 to 10.6]
Statistical Analysis 6: Comparison: LA3A (Men ACWY-CRM + Infant Vaccines) vs LA3B (Men ACWY-CRM + Infant Vaccines); Hib (≥ 0.15 μg/mL) (percentage difference (LA3A - LA3B)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 41, analysis 1]; ANOVA; Percentage difference = 0, 95% CI 2-sided [-3.1 to 3.6]
Statistical Analysis 7: Comparison: LA3A (Men ACWY-CRM + Infant Vaccines) vs LA3B (Men ACWY-CRM + Infant Vaccines); Hib (≥1.0 μg/mL) (percentage difference (LA3A - LA3B)); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 41, analysis 1]; ANOVA; Percentage difference = 1, 95% CI 2-sided [-2.2 to 5.3]

42. Secondary Outcome: Percentage of Subjects With hSBA ≥1:8 at 1 Month After 1st (LA2) or 2nd (LA4) Toddler MenACWY Vaccination - LA Subjects
Description: Immunogenicity as measured by the percentage of subjects with serum bactericidal activity using human complement (hSBA) ≥ 1:8, directed against N.meningitidis serogroups A, C, W and Y.
Time Frame: 12 or 15 months of age (one month post 1st or 2nd toddler vaccination)
Population: The analysis was done on per protocol population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | LA2 (Infant Vaccines Only) | LA4 (Infant Vaccines Only)
Number analyzed (Participants) | 78 | 102
Percentages of subjects
  A Pre-vaccination (78, 101) | 0 [0 to 5] | 0 [0 to 4]
  A Post-vaccination ((78, 101) | 74 [63 to 84] | 97 [92 to 99]
  C Pre-vaccination (78, 102) | 4 [1 to 11] | 1 [0.025 to 5]
  C Post-vaccination (78, 102) | 91 [82 to 96] | 100 [96 to 100]
  W Pre-vaccination (70, 98) | 4 [1 to 12] | 5 [2 to 12]
  W Post-vaccination (70, 98) | 79 [67 to 87] | 100 [96 to 100]
  Y Pre-vaccination (71, 95) | 3 [0 to 10] | 0 [0 to 4]
  Y Post-vaccination (71, 95) | 72 [60 to 82] | 100 [96 to 100]

43. Secondary Outcome: Geometric Mean hSBA Titers at 1 Month After 1st (LA2) or 2nd (LA4) Toddler MenACWY Vaccination - LA Subjects
Description: as for outcome 35
Time Frame: 12 or 15 months of age (one month post 1st or 2nd toddler vaccination)
Population: The analysis was done on per protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | LA2 (Infant Vaccines Only) | LA4 (Infant Vaccines Only)
Number analyzed (Participants) | 78 | 108
Titers
  A Pre-vaccination (78, 101) | 2.02 [1.7 to 2.4] | 2.02 [1.74 to 2.35]
  A Post-vaccination (78, 101) | 25 [18 to 34] | 128 [97 to 169]
  C Pre-vaccination (78, 102) | 2.18 [1.73 to 2.74] | 2.05 [1.68 to 2.51]
  C Post-vaccination (78, 102) | 45 [34 to 60] | 501 [391 to 643]
  W Pre-vaccination (70, 98) | 2.34 [1.79 to 3.05] | 2.33 [1.86 to 2.91]
  W Post-vaccination (70, 98) | 22 [16 to 28] | 394 [313 to 497]
  Y Pre-vaccination (71, 95) | 2.2 [1.7 to 2.84] | 2.04 [1.64 to 2.55]
  Y Post-vaccination (71, 95) | 15 [11 to 20] | 329 [254 to 426]

ADVERSE EVENTS:
Groups:
- US1+US3: Groups MenACWY-CRM + Infant Vaccines (US1 +US3) pooled. US infants received MenACWY at 2, 4 and 6 months of age along with routine infant vaccines, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccine. These infants either received a fourth dose of MenACWY concomitantly with pneumococcal, HAV, and MMR-V vaccines at 12 months of age (US1A and US3) or received pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months and a fourth dose of MenACWY at 13 months of age( US1B).
- US2+US4A+US4B: Groups Infant Vaccines only (US2, US4A, and US4B) pooled.
  In both groups US infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. These infants received:
  1. One dose of MenACWY concomitantly with pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and a second dose of MenACWY at 15 months of age ( US2 and US4A).
  2. Concomitant pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months and one dose of MenACWY at 13 and a second dose of MenACWY at 15 months of age (US4B)
- US4C: US infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines, at 2, 4 and 6 months of age. These subjects received concomitant pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months and one dose of MenACWY at 18 months of age.
- LA1+LA3+LA5: Groups Men ACWY-CRM + Infant Vaccines (LA1, LA3 and LA5) pooled
  LA infants received MenACWY at 2 and 6 months of age; and DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. These infants received at 12 months of age pneumococcal conjugate vaccine, HAV, and MMR-V and concomitant third dose of MenACWY (LA1A) or a third dose of MenACWY at 13 months of age (LA1B).
  LA infants received MenACWY, DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. At 12 months of age these infants received pneumococcal conjugate vaccine, HAV, and MMR-V and received:
  1. Fourth dose of MenACWY concomitantly with DTaP and Hib at 16 months of age (LA3A)
  2. DTaP and Hib at 16 months and fourth dose of MenACWY at 17 months of age (LA3B).
  3. Concomitantly the fourth dose of MenACWY (LA5).
- LA2+4+6AB: Groups Infant Vaccines only (LA2, LA4, LA6A and LA6B) pooled. In all groups LA infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus and pneumococcal conjugate vaccines at 2, 4 and 6 months of age. These infants either received: one dose of MenACWY concomitantly with pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months and a second dose of MenACWY at 15 months of age (LA2 and LA4) or received concomitant pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months and one dose each of MenACWY at 12 and 15 months of age (LA6A); or one dose each of MenACWY at 13 and 15 months of age (LA6B).
- LA6C: LA infants received as part of routine infant vaccination schedule DTaP-IPV-HBV, Hib, rotavirus, and pneumococcal conjugate vaccines, at 2, 4 and 6 months of age. These infants received concomitant pneumococcal conjugate vaccine, HAV, and MMR-V at 12 months; and one dose of MenACWY at 18 months of age
Arm/Group | US1+US3 | US2+US4A+US4B | US4C | LA1+LA3+LA5 | LA2+4+6AB | LA6C
Serious Adverse Events (participants affected / at risk) | 58/995 | 18/301 | 14/203 | 173/2026 | 84/824 | 12/183
Other Adverse Events (participants affected / at risk) | 957/995 | 279/301 | 202/203 | 1946/2026 | 795/824 | 178/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | US1+US3 (N=995) | US2+US4A+US4B (N=301) | US4C (N=203) | LA1+LA3+LA5 (N=2026) | LA2+4+6AB (N=824) | LA6C (N=183)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
LYMPHADENITIS (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
CYANOSIS (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0
PULMONARY VALVE STENOSIS (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
FALLOT'S TETRALOGY (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
HYPOSPADIAS (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
OPTIC NERVE HYPOPLASIA (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0
PYLORIC STENOSIS (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0
HAEMATOTYMPANUM (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
BLEPHARITIS (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 0 | 8 | 4 | 0
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
INTUSSUSCEPTION (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
PERITONITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
VOMITING (Gastrointestinal disorders) | 1 | 1 | 0 | 4 | 3 | 1
OEDEMA (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
PYREXIA (General disorders) | 3 | 0 | 0 | 5 | 5 | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 | 0 | 0 | 1 | 0 | 0
FOOD ALLERGY (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
ABSCESS LIMB (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0
ABSCESS NECK (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
ABSCESS ORAL (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
ACARODERMATITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
ACUTE SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
ARTHRITIS BACTERIAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
BACTERAEMIA (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
BACTERIAL DIARRHOEA (Infections and infestations) | 0 | 0 | 0 | 3 | 6 | 0
BOTULISM (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
BRONCHIOLITIS (Infections and infestations) | 10 | 3 | 2 | 32 | 16 | 6
BRONCHITIS (Infections and infestations) | 0 | 0 | 0 | 6 | 1 | 2
BRONCHITIS VIRAL (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
CELLULITIS (Infections and infestations) | 3 | 0 | 0 | 0 | 1 | 1
CROUP INFECTIOUS (Infections and infestations) | 1 | 0 | 1 | 3 | 0 | 0
DENGUE FEVER (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0
ENTERITIS INFECTIOUS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
EXANTHEMA SUBITUM (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
FEBRILE INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 2 | 0 | 2 | 14 | 4 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
IMPETIGO (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
INFECTIOUS MONONUCLEOSIS (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
INFLUENZA (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
LUNG INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
OSTEOMYELITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
OTITIS MEDIA (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 0
OTITIS MEDIA ACUTE (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
PERIORBITAL CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 2 | 2 | 0
PERTUSSIS (Infections and infestations) | 1 | 0 | 0 | 2 | 2 | 0
PHARYNGITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 4 | 2 | 1 | 37 | 9 | 2
PNEUMONIA BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 5 | 2 | 0
PNEUMONIA PRIMARY ATYPICAL (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
PNEUMONIA RESPIRATORY SYNCYTIAL VIRAL (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
PNEUMONIA VIRAL (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0
RESPIRATORY SYNCYTIAL VIRUS BRONCHIOLITIS (Infections and infestations) | 4 | 4 | 1 | 0 | 0 | 1
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 3 | 0 | 0 | 2 | 0 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
SEPSIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
STAPHYLOCOCCAL ABSCESS (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
STAPHYLOCOCCAL SKIN INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 | 0 | 1 | 4 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 1 | 0 | 9 | 8 | 0
VARICELLA (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
VIRAL DIARRHOEA (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
VIRAL INFECTION (Infections and infestations) | 1 | 0 | 1 | 1 | 2 | 0
VIRAL PHARYNGITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
VULVAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
ACCIDENTAL DRUG INTAKE BY CHILD (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
ACCIDENTAL EXPOSURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
BURNS SECOND DEGREE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
FOREIGN BODY (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0
LIMB TRAUMATIC AMPUTATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
SKULL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 0 | 0
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2 | 0 | 0
TRAUMATIC BRAIN INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
COW'S MILK INTOLERANCE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 5 | 1 | 2 | 1 | 1 | 2
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
SYNOSTOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
COMPLEX PARTIAL SEIZURES (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
CONVULSION (Nervous system disorders) | 2 | 1 | 0 | 5 | 0 | 0
FEBRILE CONVULSION (Nervous system disorders) | 1 | 0 | 1 | 13 | 4 | 1
GRAND MAL CONVULSION (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
PSYCHOMOTOR SKILLS IMPAIRED (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
TONIC CONVULSION (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
NEPHROTIC SYNDROME (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
APNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 6 | 3 | 0
BRONCHIAL HYPERREACTIVITY (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5 | 2 | 1
CHOKING (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
FOREIGN BODY ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
LARYNGOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
STATUS ASTHMATICUS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
INTESTINAL OPERATION (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
KAWASAKI'S DISEASE (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | US1+US3 (N=995) | US2+US4A+US4B (N=301) | US4C (N=203) | LA1+LA3+LA5 (N=2026) | LA2+4+6AB (N=824) | LA6C (N=183)
CONJUNCTIVITIS (Eye disorders) | 93 | 30 | 29 | 68 | 28 | 9
DIARRHOEA (Gastrointestinal disorders) | 289 | 91 | 78 | 597 | 287 | 57
FLATULENCE (Gastrointestinal disorders) | 23 | 8 | 12 | 0 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 49 | 11 | 12 | 53 | 29 | 1
TEETHING (Gastrointestinal disorders) | 83 | 28 | 30 | 11 | 2 | 0
VOMITING (Gastrointestinal disorders) | 217 | 69 | 61 | 486 | 228 | 39
INJECTION SITE ERYTHEMA (General disorders) | 280 | 108 | 100 | 1245 | 548 | 117
INJECTION SITE INDURATION (General disorders) | 204 | 101 | 78 | 745 | 333 | 90
INJECTION SITE PAIN (General disorders) | 651 | 196 | 147 | 1592 | 698 | 164
IRRITABILITY (General disorders) | 800 | 240 | 171 | 1120 | 474 | 110
MALAISE (General disorders) | 0 | 0 | 0 | 136 | 73 | 5
PYREXIA (General disorders) | 296 | 94 | 74 | 748 | 341 | 74
BRONCHIOLITIS (Infections and infestations) | 108 | 34 | 25 | 180 | 52 | 36
BRONCHITIS (Infections and infestations) | 10 | 6 | 5 | 219 | 95 | 17
CROUP INFECTIOUS (Infections and infestations) | 44 | 12 | 15 | 2 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 49 | 18 | 6 | 48 | 35 | 3
NASOPHARYNGITIS (Infections and infestations) | 41 | 9 | 11 | 375 | 192 | 27
OTITIS MEDIA (Infections and infestations) | 258 | 76 | 62 | 26 | 17 | 2
OTITIS MEDIA ACUTE (Infections and infestations) | 42 | 15 | 13 | 37 | 15 | 7
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0 | 0 | 163 | 71 | 5
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 340 | 108 | 74 | 16 | 4 | 0
VIRAL INFECTION (Infections and infestations) | 82 | 22 | 20 | 44 | 28 | 1
CRYING (Nervous system disorders) | 558 | 154 | 124 | 927 | 419 | 98
SOMNOLENCE (Nervous system disorders) | 676 | 184 | 141 | 1198 | 513 | 110
EATING DISORDERS (Psychiatric disorders) | 425 | 122 | 93 | 607 | 263 | 69
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 15 | 0 | 3 | 38 | 7 | 15
COUGH (Respiratory, thoracic and mediastinal disorders) | 64 | 20 | 15 | 41 | 24 | 4
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 60 | 15 | 18 | 6 | 1 | 1
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 29 | 9 | 13 | 26 | 16 | 1
DERMATITIS DIAPER (Skin and subcutaneous tissue disorders) | 62 | 21 | 13 | 8 | 4 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 105 | 32 | 21 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 154 | 33 | 39 | 323 | 136 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days